

Statistical Analysis Plan

Protocol No: 20130108

10-December-2018/ Version 2.0

# **Statistical Analysis Plan**

A Randomized, Double-Blind Study to Compare Pharmacokinetics and Pharmacodynamics, Efficacy and Safety of ABP 798 with Rituximab in Subjects with Moderate to Severe Rheumatoid Arthritis

| Sponsor: | Amgen Inc. |
|-----------------|---------------------------------------------|
| Protocol No: | 20130108 - Date 20-March-2018 - Version 4.0 |
| PRA Project Id: | AMGRA798-798RAX |
| Version Date: | 10-December-2018 |
| Version Number: | 2.0 |

# APPROVALS

| Sponsor Name: | Amgen Inc. |
|---|---|
| Name of Sponsor<br>Representative/Title: | / Clinical Research Medical Director, Amgen Inc. |
| Signature of Sponsor<br>Representative /Date: | 10 DEC2018 |
| Name of Sponsor<br>Representative/Title: | PPD // Biostatistics Sr. Manager, Amgen Inc. |
| Signature of Sponsor<br>Representative /Date: | 10 Dec 2018 |
| Name of Project<br>Manager/Title: | / Project Manager |
| Signature of Project<br>Manager/Date: | 10 Dec 2018 |
| Name of<br>Biostatistician /Title: | PPD / Principal Biostatistician |
| Signature of<br>Biostatistician /Date: | PPD 10 10 (2012<br>FOR PPD |
| | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |

(NOTE: Electronic Signatures should only be used if all parties have the ability to eSign.)



# Statistical Analysis Plan

10-December-2018/ Version 2.0

Protocol No: 20130108

# TABLE OF CONTENTS

| Approvals | 1 |
|--------------------------------------------------------------|----|
| Table of Contents | 2 |
| 1. Introduction | 6 |
| 2. Study Objectives | 6 |
| 2.1 Primary Objectives | 6 |
| 2.2 Secondary Objectives | 6 |
| 3. Study Design | 6 |
| 3.1 Sample Size Considerations | 8 |
| 3.2 Randomization | 9 |
| 4. Study Variables and Covariates | 9 |
| 4.1 Primary Variable | 9 |
| 4.2 Secondary Variables | 9 |
| 4.2.1 Pharmacokinetic | 9 |
| 4.2.2 Efficacy | 10 |
| 4.2.3 Pharmacodynamic | 10 |
| 4.2.4 Safety | 10 |
| 4.3 Predetermined Covariates and Prognostic Factors | 10 |
| 5. Definitions | 11 |
| 5.1 General | 11 |
| Actual Treatment Received | 11 |
| Baseline | 12 |
| Binding and Neutralizing ADA status During First Dose Period | 12 |
| Change from Baseline | 12 |
| Completed Study | 12 |
| Concomitant and Prior Medication | 13 |
| Duration of IP Exposure | 13 |
| Early Retreatment | 13 |
| End of Study Date | 13 |
| First Dose Date | 13 |
| Infusion delay | 13 |
| Infusion missed | 13 |
| Last Dose Date | 13 |
| Percent Improvement from Baseline | 14 |
| RA Disease Duration | 14 |
| Seropositivity | 14 |
| Study Day 1 | 14 |



# Statistical Analysis Plan

Protocol No: 20130108

10-December-2018/ Version 2.0

| | Stı | udy Day | 14 |
|---|---|---|---|
| | Stı | udy Randomization | 15 |
| | Stı | udy Visit | 15 |
| | | For PK analyses: | 15 |
| | | For efficacy analyses: | |
| | | For safety (Hematology and chemistry) analyses: | 17 |
| | | For CD19+, IgA, IgM and IgG analysis: | 17 |
| | | For vital signs analyses: | 17 |
| | | For ADA analyses: | 18 |
| | 5.2 | Pharmacokinetic | |
| | 5.3 | Efficacy | 20 |
| | A( | CR20/50/70 | 20 |
| | DA | AS28-CRP | 20 |
| | DA | AS28-CRP Remission | 21 |
| | Не | ealth Assessment Questionnaire – Disability Index (HAQ-DI) | 21 |
| | Ну | ybrid ACR Response | 21 |
| | Sv | vollen Joint Count | 21 |
| | Te | ender Joint Count | 21 |
| | 5.4 | Safety | 22 |
| | Ac | dverse Event of Interest (AEOI) | 22 |
| | | sposure Adjusted Incidence Rate (EAIR) for Adverse Events and Adverset 22 | erse Event of |
| | Su | bject Incidence Rate | 23 |
| | Tr | reatment-emergent Adverse Event | 23 |
| | 5.5 | PHARMACODYNAMICS | 23 |
| | Co | omplete depletion of CD19+ cell count | 23 |
| | Dι | uration of CD19+ B-cell complete depletion | 23 |
| 6. | Ar | nalysis Sets | 23 |
| | 6.1 | Full Analysis Set | 23 |
| | 6.2 | Per-protocol Analysis Set | 24 |
| | 6.3 | Safety Analysis Set | 24 |
| | 6.4 | Pharmacokinetic Concentration Analysis Set | 24 |
| | 6.5 | Pharmacokinetic Parameter Analysis Set | 24 |
| | 6.6 | Per-protocol Pharmacokinetic Parameter Analysis Set | 24 |
| | 6.7 | Anti-drug Antibody Analysis Set | 25 |
| <b>7.</b> | In | terim Analyses | 25 |
| 8. | Da | ata Review | 25 |
| | 8 1 | Data Handling and Transfer | 25 |



# Statistical Analysis Plan

Protocol No: 20130108 10-December-2018/ Version 2.0

| 8.2 | 2 D | ata Screening | 26 |
|---|---|---|---|
| 9. | Statist | ical Methods | 26 |
| 9. | 1 Su | ubject Disposition | 26 |
| 9.2 | 2 Pr | rotocol Deviations | 27 |
| 9 | 3 T <sub>1</sub> | reatments | 27 |
| | 9.3.1 | Extent of IP Exposure | 27 |
| | 9.3.2 | Prior and Concomitant Medications | 27 |
| 9.4 | 4 D | emographic and Baseline Characteristics | 28 |
| 9.: | 5 Pl | narmacokinetic analyses | 29 |
| | 9.5.1 | Pharmacokinetic Concentrations | 29 |
| | 9.5.2 | Pharmacokinetic Parameters | 29 |
| | Prin | nary Statistical Analysis | 30 |
| | Sens | sitivity Analyses | 30 |
| 9. | 6 Pł | narmacodynamics Analyses | 31 |
| | 9.6.1 | CD19 | 31 |
| | 9.6.2 | IgA, IgG and IgM | 31 |
| 9. | 7 E | fficacy Analyses | 31 |
| | 9.7.1 | DAS28-CRP. | 32 |
| | Prin | nary StatisTical Analysis | 32 |
| | Sens | sitivity Analyses | 33 |
| | 9.7.2 | ACR 20/50/70 | |
| | 9.7.3 | Hybrid ACR | |
| | 9.7.4 | Methods for Handling Dropouts and Missing Data for Efficacy | |
| | 9.7.5 | Multiplicity | |
| | 9.7.6 | Pooling of Sites | |
| 9. | | afety Analyses | |
| | 9.8.1 | Adverse Events | |
| | 9.8.2 | Deaths and Serious Adverse Events | |
| | 9.8.3 | Laboratory Data | |
| | 9.8.4 | Vital Signs and Physical Examination | |
| | 9.8.5 | Immunogenicity | |
| | 9.8.6 | Methods for Handling Missing Data for Safety | |
| 9.9 | | xploratory Analyses | |
| | 9.9.1 | DAS28-CRP Individual Components | |
| | 9.9.2 | ACR Individual Components | |
| 10. | | ANGE FROM PROTOCOL SPECIFIED ANALYSIS | |
| 11. | Vali | dation | 42 |



| Sponsor: An | mgen Inc. Statistica | Statistical Analysis Plan |
|---|---|---|
| Protocol No: | : 20130108 10-December-2 | 10-December-2018/ Version 2.0 |
| 12. Refere | rences | 42 |
| Appendix 1 | Glossary of Abbreviations | 43 |
| Appendix 2 | Method for missing individual components of ACR ca | alculation46 |
| Appendix 3 | Method for Missing individual joint assessments | 47 |
| Appendix 4 | HAQ-DI Scoring Algortihm | 49 |
| • • | List of Events of Interest and the Associated SMQ and I | U |
| Appendix 6 | List of Post-Text Tables, Figures, Listings, and Suppo | ortive SAS |
| <b>Output App</b> | pendices | 52 |
| Appendix 7 | Shells for Post-Text Tables, Figures, and Listings | 73 |




# 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical methods to be used during the reporting and analyses of data collected under Amgen Inc. Protocol 20130108, titled "A Randomized, Double-Blind Study to Compare Pharmacokinetics and Pharmacodynamics, Efficacy and Safety of ABP 798 with Rituximab in Subjects with Moderate to Severe Rheumatoid Arthritis."

This SAP should be read in conjunction with the study protocol and electronic Case Report Forms (eCRFs). This version of the plan has been developed using the protocol version 4.0 dated 20 March 2018 and eCRFs version 5.0 dated 17 November 2016. Any further changes to the protocol or eCRFs may necessitate updates to the SAP.

The SAP is to be developed in two stages. The purpose is to "finalize" a SAP in order to start programming earlier in the process. Versions of the SAP up to initial sponsor approval will be known as SAP1. Changes following approval of SAP1will be tracked in the SAP Change Log and a final version of the SAP, known as SAP2, will be issued for Amgen's approval prior to unblinding for the final analysis.

# 2. STUDY OBJECTIVES

#### 2.1 PRIMARY OBJECTIVES

The primary objective for this study is to demonstrate pharmacokinetic (PK) similarity (as assessed principally by area under the serum concentration-time curve [AUC] from time 0 extrapolated to infinity [AUC $_{inf}$ ] and the maximum observed serum concentration [C $_{max}$ ], following the 2nd infusion of the 1st dose) of ABP 798 following 2 intravenous (IV) infusions of 1000 mg each, relative to that of 2 IV infusions of 1000 mg each of rituximab (US) and of rituximab (EU).

#### 2.2 SECONDARY OBJECTIVES

The secondary objectives are:

- to demonstrate PK similarity between rituximab (US) and rituximab (EU) as assessed by AUC<sub>inf</sub> and by C<sub>max</sub> after second infusion of the first dose
- to assess the clinical efficacy of ABP 798 compared with rituximab
- to assess the safety and immunogenicity of ABP 798 compared with rituximab.

# 3. STUDY DESIGN

This is a randomized, double-blind, active-controlled 3-arm study in adult subjects with moderate to severe Rheumatoid Arthritis (RA) who have an inadequate response or intolerance to other disease-modifying anti-rheumatic drugs (DMARDs), which must include intolerance or inadequate response to one or more tumor necrosis factor (TNF) inhibitor therapies.




Approximately 300 subjects (100 per treatment group) will be enrolled. The subjects will be randomized to receive either 2 IV infusions of ABP 798, 1000 mg each, given 2 weeks apart (treatment group A), or 2 IV infusions of rituximab (US) 1000 mg each, given 2 weeks apart (treatment group B) or 2 IV infusions of rituximab (EU), 1000 mg each, given 2 weeks apart (treatment group C) in a double blind fashion. A total of 2 doses will be administered during the study; each dose consists of 2 infusions, 2 weeks apart.

An independent data monitoring committee (DMC) will evaluate the safety data throughout the study, including an initial safety analysis after the first 18 subjects have received the first dose (1000 mg x 2 infusions of either ABP 798 or rituximab (EU) or rituximab (US)).

At week 24, the subjects in treatment groups A and C will continue with and receive the second dose of the same treatment, and the subjects in treatment group B will transition to treatment group A1 and receive ABP 798 1000 mg x 2 as their second dose. Retreatment may occur earlier, i.e., anytime from week 16 to week 24, in individual subjects, if necessary in the opinion of the Investigator.

The end of study (EOS) will be at week 48 (or 24 weeks after the first infusion of second dose for subjects retreated before week 24), and a final analysis will be performed when all subjects have completed or have had the opportunity to complete the week 48/EOS assessments.

See Figure 1 below for a summary of the study design.


Figure 1 **Study Diagram** 



<sup>\*</sup> Retreatment will begin at week 24 or earlier, i.e., anytime from week 16 to week 24 in individual subjects if necessary in the opinion of the Investigator.

# SAMPLE SIZE CONSIDERATIONS

Approximately 300 subjects will be randomized in a 1:1:1 ratio to receive ABP 798, rituximab (US), or rituximab (EU), stratified by geographic region (North America, Eastern Europe, and Western Europe), seropositivity (rheumatoid factor (RF)-positive and/or anti-cyclic citrullinated peptide (CCP)-positive vs. RF-negative and CCPnegative), and number of prior biologic therapies used for RA (1 vs. >1). The sample size will provide > 90% power to demonstrate similarity on the primary PK endpoints based on an assumption of between-subject variability (as measured by coefficient of variation) of 40%, true geometric mean ratio (GMR) of 1 among ABP 798, rituximab (US), or rituximab (EU), a margin of (0.8, 1.25) and 15% dropout by week 24. PK similarity will


be tested between ABP 798 versus rituximab (US) and ABP 798 versus rituximab (EU), each with a significance level of 0.05. The similarity between rituximab (US) and rituximab (EU) will be evaluated as well.

With the planned sample size, there is 94% probability that the 90% CI of the difference between the ABP 798 arm and the pooled rituximab (rituximab [EU] and rituximab [US]) arm and 83% probability that the 90% CI of the difference between test (ABP 798) and reference (rituximab [EU] or rituximab [US]) in DAS28-CRP change from baseline at week 24 will fall into the equivalence margin of  $\pm 0.6$  (EULAR response criteria), assuming a standard deviation of 1.4 (Volkmann et al. 2010) and true mean difference of 0.

# 3.2 RANDOMIZATION

Approximately 300 subjects will be randomized in a 1:1:1 ratio to receive either ABP 798, rituximab (US), or rituximab (EU) via an Interactive Voice or Web Response System (IXRS), stratified by geographic region (North America, Eastern Europe, and Western Europe), seropositivity (RF-positive and/or CCP-positive vs. RF-negative and CCPnegative), and number of prior biologic therapies used for RA (1 vs. >1).

Assignment to the treatment arms will be based on a computer-generated randomization schedule created before the start of the study. The randomization schedule will be prepared by a statistician not involved in the conduct of the study.

A third party vendor, , will be responsible for generating the randomization scheme and managing the randomization activities of this study.

#### 4. STUDY VARIABLES AND COVARIATES

# 4.1 PRIMARY VARIABLE

The primary PK endpoints are the AUC<sub>inf</sub> and C<sub>max</sub> following the 2<sup>nd</sup> infusion of 1<sup>st</sup> dose.

# 4.2 SECONDARY VARIABLES

#### 4.2.1 Pharmacokinetic

The secondary PK endpoints will include:

- AUC from time 0 on day 1 prior to the 1<sup>st</sup> infusion of the 1<sup>st</sup> dose to 14 days postdose (AUC<sub>0-14 day</sub>)
- AUC from time 0 on day 1 prior to the 1<sup>st</sup> infusion of the 1<sup>st</sup> dose to week 12  $(AUC_{0-12 \text{ wk}})$
- C<sub>max</sub> following the 1<sup>st</sup> infusion of the 1<sup>st</sup> dose.


Additional PK endpoints including the time of  $C_{max}$  ( $t_{max}$ ), last measurable serum concentration after the second infusion up to week 12 (Clast), terminal elimination half-life ( $t_{1/2}$ ), the terminal elimination rate constant ( $\lambda_z$ ), clearance (CL), mean residence time (MRT), percent of AUC extrapolation (%AUC<sub>extrap</sub>), and AUC<sub>0-12</sub> wk/AUCinf.

# 4.2.2 Efficacy

The efficacy endpoints include:

Primary efficacy endpoint:

• Disease activity score (DAS) 28-CRP change from baseline at week 24.

Secondary efficacy endpoints:

- DAS 28-CRP change from baseline at week 8, 12, 40 and 48.
- ACR20, ACR50 and ACR70 at weeks 8, 12, 24, 40 and 48.
- Hybrid ACR at weeks 8, 12, 24, 40 and 48.

# 4.2.3 Pharmacodynamic

Pharmacodynamic (PD) endpoints will include the percent of subjects with complete depletion in CD19+ cell count from day 1 to day 3 and duration of CD19+ B-cell complete depletion.

# **4.2.4 Safety**

Safety endpoints include the following:

- Treatment-emergent adverse events (TEAE) and serious adverse events (SAE).
- Clinically significant changes in laboratory values.
- Changes in vital signs.
- Incidence of anti-drug antibodies.

# 4.3 PREDETERMINED COVARIATES AND PROGNOSTIC FACTORS

For the PK analyses, geographic region and weight will be used as covariates in the model for the primary statistical analysis. The following covariates may be used for further exploration in subgroups:

- Negative binding anti-drug antibodies (ADA) during first dose period
- Negative neutralizing ADA during first dose period

For efficacy analyses, unless stated otherwise, the following stratification factors will be included as covariates in the model or be used to examine treatment effect in subgroups:

Geographic region (North America vs. Eastern Europe vs. Western Europe)


Seropositivity (RF-positive and/or CCP-positive vs. RF-negative and CCP-negative)

• Prior biologic use for RA (1 vs >1)

In case the analysis model doesn't converge, the strata with least number of subjects may be combined to address the convergence issues.

In addition, the following covariates may be used for further exploration in subgroups or as covariates:

- Age Group (<65 years vs  $\ge 65$  years)
- Race (Caucasian vs Non-Caucasian)
- Gender
- Binding ADA status during first dose period (negative vs positive)
- Neutralizing ADA status during first dose period (negative vs positive)
- Oral Corticosteroid use at baseline (Yes vs No)

Additional baseline demographic and disease characteristics in Section 9.4 may also be considered as covariates in the model for assessing DAS28-CRP change from baseline at week 24.

Analyses that are intended to evaluate the treatment effect and include stratification variables as covariates in the model will be based on the eCRF stratification values, regardless of the subject's IXRS stratification values, to provide unbiased estimates of the effects of treatment and stratification variables without loss of efficiency (Ke et al, 2017).

For subgroup analyses where the subgroup factor is a stratification variable, an analysis similar to the primary statistical analysis (except the inclusion of the subgroup factor) should be done for each subgroup defined by the eCRF values of the subgroup factor.

#### 5. DEFINITIONS

# 5.1 GENERAL

# **Actual Treatment Received**

The actual treatment received is the investigational product (IP) treatment the subject actually received, regardless of what the subject was randomized to. In cases where a subject received more than 1 IP during a dose, the actual treatment received for that dose will be based on the first IP infusion of the dose the subject received. The actual treatment received for the entire study will be based on the combination of the actual treatment received for the first infusion of the two doses. In cases where a subject received only the 1<sup>st</sup> dose of IP, the actual treatment received for the entire study will be determined by the actual treatment of the 1<sup>st</sup> IP dose and the intended treatment of the 2<sup>nd</sup>


dose per protocol. The actual treatment for the study will be unplanned if the sequence of the actual treatment of each dose are not described in the protocol.

Specifically, by design for each subject, 2 doses will be administered during the study where each dose consists of 2 infusions, and each infusion consists of 2 boxes. In the cases where a subject receives mismatched boxes (differing IP) among the 2 possible boxes within an infusion, if either box is ABP 798 then the actual treatment for the infusion will be ABP 798.

#### Baseline

For the endpoint of interest, the baseline is defined as the last non-missing assessment taken prior to the first infusion of the first dose of study IP. In cases where baseline assessments are taken on the same day as the first infusion of the first dose of IP, and either no times are reported or the IP and assessment times are the same, it will be assumed that these assessments are taken prior to IP being administered. For subjects who are randomized but not dosed after the randomization, the baseline is defined as the last non-missing assessment prior to or on the date of randomization.

For the ADA analysis following the 1<sup>st</sup> infusion of the 2<sup>nd</sup> dose, the baseline is defined as last non-missing assessment prior to the 1<sup>st</sup> infusion of the 2<sup>nd</sup> dose.

# Binding and Neutralizing ADA status During First Dose Period

Subjects will be considered to have negative binding ADA status during first dose period if subjects had negative binding ADA

- from baseline up to 1st infusion of 2nd dose for subjects who received 2nd dose, or
- from baseline up to week 24 (day 175) or EOS (whichever is earlier) for subjects who didn't receive 2<sup>nd</sup> dose.

Subjects will be considered to have positive binding ADA status during first dose period if subjects had positive binding ADA status at any time point

- up to the 1<sup>st</sup> infusion of the 2<sup>nd</sup> dose for subjects who received 2<sup>nd</sup> dose, or
- up to week 24 (day 175) or EOS (whichever is earlier) for subjects who didn't receive 2<sup>nd</sup> dose.

The same definition applies to subjects' neutralizing ADA status. Subjects with a binding negative or no result at baseline and at least one post baseline will be included in this derivation.

# **Change from Baseline**

Change from baseline is defined as (value at post-baseline visit – value at baseline).

#### **Completed Study**

A subject is considered to have completed the study if they indicated they completed study on the EOS eCRF.




# **Concomitant and Prior Medication**

Prior medications are defined as medications with a stop date prior to the first infusion of the first dose of study IP. Concomitant medications are defined as any medications ongoing at the start of IP treatment or with a start date on or after the first dose date.

# **Duration of IP Exposure**

For subjects who received 2<sup>nd</sup> dose of IP, the duration of IP exposure will be derived as min (EOS date, analysis data cutoff date) minus date of first IP exposure + 1 day.

For subjects who didn't receive 2<sup>nd</sup> dose of IP, the duration of IP exposure will be derived as min (EOS date, week 24 [day 175], analysis data cutoff date) minus date of first IP exposure + 1 day.

#### **Early Retreatment**

If 1st infusion of 2nd dose is administered prior to Study Day 162, subjects are considered as receiving early retreatment.

# **End of Study Date**

EOS date is the date recorded on the End of Study page of the eCRF for a randomized subject.

# First Dose Date

The date on which a subject is administered the first infusion of first dose of study IP. This date is also referred to as Study Day 1.

#### **Infusion delay**

If an IP administration form for a visit is entered with an infusion administered of NONE and a reason for delay/not administered, and also there is infusion information entered on a subsequent IP form, that subject is considered having an infusion delay.

There is one exception. If the second infusion of the 1st dose is delayed for such a large extended period that it falls at week 16 or after, the infusion will be entered in the week 24 folder. In this case, the Day 15 IP infusion will be considered missing instead of delayed.

# **Infusion missed**

When a subject with an IP administration form entering an infusion administered of NONE and a reason for delay/not administered but there is no subsequent IP form with infusion information, the subject is considered to have missed an infusion at that visit.

In addition, if the second infusion of the 1st dose is delayed for such a large extended period that it falls at week 16 or after, the infusion will be entered in the week 24 folder. In this case, the Day 15 IP infusion will be considered missing.

#### **Last Dose Date**

The date on which a subject is administered the last infusion of the last dose of study IP.




# **Percent Improvement from Baseline**

For endpoints where higher scores indicate greater severity, the percent improvement from baseline is: (value at baseline – value at post-baseline visit) X 100 / (value at baseline).

For endpoints where lower scores indicate greater severity, the percent improvement from baseline is: (value at post-baseline visit – value at baseline) X 100 / (value at baseline).

If the baseline value is 0 and the post-baseline value is also 0, then the percent improvement from baseline is set to 0. If the baseline value is 0 and the post-baseline value is non-zero, then the percent improvement from baseline is set to "missing" (or '.').

# **RA Disease Duration**

The RA disease duration is the number of years from the date of diagnosis of RA to the date of randomization, which will be derived based on the table below. No imputation will be done for disease diagnosis date, but to avoid a disease duration of zero, 1 month (or 1/12 years) may be added.

Table 1 Calculation of the Duration of RA

| Observed | Missing | Formula to Calculate Duration |
|--------------|---------|-------------------------------------------------|
| portion | portion | |
| Year, Month, | | (Date of Randomization – Date of RA Diagnosis + |
| Day | | 1)/365.25 |
| Year, Month | Day | [Year(Date of Randomization)-Year(Date of RA |
| | _ | Diagnosis)]+ [Month(Date of Randomization)- |
| | | Month(Date of RA Diagnosis)]/12* |
| Year | Month, | [Year(Date of Randomization)-Year(Date of RA |
| | Day | Diagnosis)] * |

<sup>\*</sup>If the duration equals 0, add 1 month or 1/12 years.

# Seropositivity

For seropositivity summary at baseline, a normal or negative baseline result for RF would be <12 IU/mL and for CCP3 would be <20 Units based on the laboratory assay maker's guidance.

# **Study Day 1**

Study Day 1 is defined as the first day of IP administration. For subjects who are randomized but not dosed after the randomization, study day 1 is defined as the date of randomization.

#### **Study Day**

Study day is defined as the number of days from Study Day 1.

• Before Study Day 1:

Statistical Analysis Plan Sponsor: Amgen Inc.


Study Day = (Date of Interest – Date of Study Day 1)

• On or After Study Day 1:

Study Day = (Date of Interest – Date of Study Day 1) + 1

Therefore the day prior to Study Day 1 is -1.

# **Study Randomization**

Study randomization is defined as when subject receives a random treatment allocation via the IXRS system.

# **Study Visit**

Since the actual visit for a subject may not exactly coincide with their scheduled visit date, the actual visit date is mapped to the study analysis visit as follows. Note that the following analytical visit windows for statistical analysis are different from the ones defined in Section 18.0 of the IXRS Business Requirement. The actual visit date is allowed to fall within specified interval of the target day.

In general, if more than one actual visit (including the unscheduled visits) falls within the same defined window, the visit closest to the target day with non-missing data will be considered for analysis. If two actual visit dates are at the same distance from the target day, the latest visit with non-missing data will be considered for analysis. For Week 24, only actual visits that occur before or on same date as first infusion of second dose should be considered.

The rules above for selecting a visit from multiple ones within the same visit window are not applicable to retest values of lab data. If the lab measurement is a retest, the retest value will be chosen.

PK concentration will be summarized by the scheduled sample visit in the protocol. For PK concentration collected in the unscheduled visits or in the early discontinuation study visit, the associated scheduled sample visit is defined as below. If multiple records are assigned to the same visit, the one closest to the reference date/time will be selected into the summary.

# FOR PK ANALYSES:

| Scheduled Sample | |
|---|---|
| Visit | Window Mapping |
| | Prior to the 1st IP infusion of 1st dose start time but on the |
| Day 1 Pre-dose | same day |
| Day 1 End of infusion | within 10 minutes of 1st infusion of 1st dose stop date/time |
| | $3 \text{ hr} \pm 10 \text{ minutes after 1st IP infusion of 1st dose stop}$ |
| Day 1 3 hours | date/time |
| | 6 hours $\pm$ 10 minutes after 1st IP infusion of 1st dose stop |
| Day 1 6 hours | date/time |




| Day 2 24 hours post- | 24 hr $\pm$ 3 hours after 1st IP infusion of 1st dose stop |
|---|---|
| dose | date/time |
| Day 3 48 hours post- | $48 \text{ hr} \pm 3 \text{ hours after 1st IP infusion of 1st dose stop}$ |
| dose | date/time |
| | Prior to the 2nd IP infusion of 1st dose start time but on the |
| Day 15 Pre-dose | same day |
| Day 15 End of infraisa | within 10 minutes of 2nd infusion of 1st does ston data/time |
| Day 15 End of infusion | within 10 minutes of 2nd infusion of 1st dose stop date/time |
| D 15 2 h | $3hr \pm 10$ minutes after 2nd IP infusion of 1st dose stop |
| Day 15 3 hours | date/time |
| D 15 ( 1 | $6hr \pm 10$ minutes after 2nd IP infusion of 1st dose stop |
| Day 15 6 hours | date/time |
| Day 16 24 hours post- | 24 hr $\pm$ 3 hours after 2nd IP infusion of 1st dose stop |
| dose | date/time |
| Day 17 48 hours post- | 48hr ± 3 hours after 2nd IP infusion of 1st dose stop |
| dose | date/time |
| XXX 1 4 | 2 wks $(14 \text{ days}) \pm 2 \text{ days}$ after the 2nd infusion of 1st dose |
| Week 4 | stop date |
| | 6 wks (14 days) $\pm$ 2 days after the 2nd infusion of 1st dose |
| Week 8 | stop date |
| | 10 wks (14 days) $\pm$ 2 days after the 2nd infusion of 1st dose |
| Week 12 | stop date |
| | Prior to the 1st IP infusion of 2nd dose start time but on the |
| Week 24 Pre-dose | same day |
| | Prior to the 2nd IP infusion of 2 <sup>nd</sup> dose start time but on the |
| Week 26 Pre-dose | same day |
| | 4 wks $(28 \text{ days}) \pm 2 \text{ days}$ from the 2nd infusion of 2nd dose |
| Week 30 | stop date |
| | 22 wks $(154 \text{ days}) \pm 2 \text{ days}$ from the 2nd infusion of 2nd |
| Week 48 | dose stop date |

# FOR EFFICACY ANALYSES:

| Study Analysis Visit | <b>Target Day</b> | Study Day | Interval (days) |
|----------------------|-------------------|-----------|-----------------|
| Baseline | 1 | <u>≤1</u> | NA |
| Week 8 | 57 | 2 - 70 | 69 |
| Week 12 | 85 | 71 - 105 | 42 |
| Week 24 | 169 | 106 - 210 | 98 |
| Week 40 | 281 | 211 - 308 | 98 |
| Week 48 | 337 | ≥309 | NA |


# FOR SAFETY (HEMATOLOGY AND CHEMISTRY) ANALYSES:

| Study Analysis | <b>Target Day</b> | Study Day | Interval (days) |
|---------------------------|-------------------|-----------|-----------------|
| <u>Visit</u> <sup>a</sup> | | | |
| Baseline <sup>b</sup> | 1 | ≤1 | NA |
| Week 2 | 15 | 2 - 16 | 15 |
| Day 17 | 17 | 17 | 1 |
| Week 4 | 29 | 18 - 42 | 25 |
| Week 8 | 57 | 43 - 105 | 70 |
| Week 24 | 169 | 106 - 175 | 63 |
| Week 26 | 183 | 176 - 196 | 21 |
| Week 30 | 211 | 197 - 245 | 49 |
| Week 40 | 281 | 246 - 308 | 63 |
| Week 48 | 337 | ≥309 | NA |

<sup>&</sup>lt;sup>a</sup> Laboratory parameters will only be included at the visits where it is scheduled for assessment in the output tables.

# FOR CD19+, IGA, IGM AND IGG ANALYSIS:

| <b>Study Analysis</b> | <b>Target Day</b> | Study Day | Interval (days) |
|---------------------------|-------------------|-----------|-----------------|
| <u>Visit</u> <sup>a</sup> | | | |
| Baseline <sup>b</sup> | 1 | ≤1 | NA |
| Day 2 | 2 | 2 | 1 |
| Day 3 | 3 | 3 | 1 |
| Week 4 | 29 | 15 - 42 | 28 |
| Week 24 | 169 | 106 - 210 | 98 |
| Week 48 | 337 | ≥309 | NA |

<sup>&</sup>lt;sup>a</sup> IgG and IgA will not be collected at Day 2 and Day 3

# FOR VITAL SIGNS ANALYSES:

| Study Analysis | <b>Target</b> | Study Day <sup>b</sup> | <u>Interval</u> |
|---|---|---|---|
| <u>Visit</u> <sup>a</sup> | <b>Day</b> | | (days) |
| Baseline | NA | Day 1 prior to infusion | NA |
| Day 1 end of | NA | Day 1 after infusion | NA |
| infusion (EOI) | | | |
| Day 1 3 hours | NA | Day 1 3 hours after EOI | NA |
| Day 1 6 hours | NA | Day 1 6 hours after EOI | NA |
| Week 2 | NA | Day 15 prior to infusion | 14 |

<sup>&</sup>lt;sup>b</sup> If a subject has lab measurements on the same day as the first infusion date of first dose but at a time after the first infusion of first dose is administered, the lab measurements will not be defined as baseline, but as Week 2 measurements.

<sup>&</sup>lt;sup>b</sup> If a subject has measurements on the same day as the first infusion date of first dose but at a time after the first infusion of first dose is administered, the measurements will not be defined as baseline, but as Day 2 measurement.




| D 17 FOI | N.T.A | D 15 C 'C' | NT A |
|----------------|-------|--------------------------|------|
| Day 15 EOI | NA | Day 15 after infusion | NA |
| Day 15 3 hours | NA | Day 15 3 hours after EOI | NA |
| Day 15 6 hours | NA | Day 15 6 hours after EOI | NA |
| Week 24 | 169 | 106 - 175 | 63 |
| Week 26 | 183 | 176 – 196 | 21 |
| Week 30 | 211 | 197 - 245 | 49 |
| Week 48 | 337 | >309 | NA |

<sup>&</sup>lt;sup>a</sup>If a visit date with multiple records, the highest value per parameter will be selected for analysis.

#### FOR ADA ANALYSES:

| Study Analysis | Target Day | Study Day | Interval (days) |
|-----------------------|------------|-----------|-----------------|
| <u>Visit</u> | | | |
| Baseline <sup>a</sup> | 1 | ≤1 | NA |
| Week 2 | 15 | 2 - 16 | 15 |
| Week 24 | 169 | 106 - 175 | 63 |
| Week 30 | 211 | 197 - 245 | 49 |
| Week 48 | 337 | ≥309 | NA |

<sup>&</sup>lt;sup>a</sup> If a subject has ADA assessments on the same day as the first infusion date of first dose but at a time after the first infusion of first dose is administered, the ADA assessments will not be defined as baseline, but as Week 2 assessments.

# 5.2 PHARMACOKINETIC

Pharmacokinetic parameters will be calculated from serum concentration-time data using noncompartmental analysis (NCA) methods using Phoenix WinNonLin® Version 6.4 or higher (Pharsight Corp, St. Louis, MO). The following PK parameters will be reported for serum rituximab and ABP 798, using actual elapsed sampling times:

| Variable | Definition |
|---|---|
| $C_{max1}$ | Maximum observed serum concentration following Dose 1 Infusion 1 |
| Cmax2 | Maximum observed serum concentration following Dose 1 Infusion 2 |
| $t_{max1}$ | Time to which the maximum serum concentration was observed following Dose 1 Infusion 1 |
| t <sub>max2</sub> | Time to which the maximum serum concentration was observed following Dose 1 Infusion 2 |
| TLST1 | Time of last quantifiable concentration following Dose 1 Infusion 1 |

<sup>&</sup>lt;sup>b</sup>Day 1 and Day 15 visit/timepoint are directly associated with infusion date/time.




CLST1 Last quantifiable concentration following Dose 1 Infusion 1

over first 14 days postdose (day 15)

AUC<sub>0-14 day</sub> Area under the serum concentration-time curve from time 0

on day 1 prior to the first infusion of the first dose to last quantifiable concentration associated with Dose 1 Infusion

1 over the first 14 days postdose (day 15)

TLST2 Time of last quantifiable concentration associated with

Dose 1 Infusion 2

CLST2 Last quantifiable concentration after Dose 1 Infusion 2

AUC<sub>0-12 wk</sub> Area under the serum concentration-time curve from time 0

on day 1 prior to the first infusion of the first dose to last

quantifiable concentration over 12-week profile

AUC<sub>inf</sub> Area under the serum concentration-time curve from time 0

on day 1 prior to the first infusion of the first dose

extrapolated to infinity; calculated as AUC<sub>last</sub> + CLST2/ $\lambda_z$ ,

where AUC<sub>last</sub> is the AUC from time 0 to the last

quantifiable concentration up to week 12 (i.e. AUC<sub>0-12 wk</sub>)

 $t_{1/2}$  Terminal elimination half-life determined from time 0 to

Week 12 profile; calculated as  $\ln(2)/\lambda_z$ 

 $\lambda_z$  Terminal elimination rate constant

CL Clearance

AUMC Area under the first moment curve

MRT Mean residence time; calculated as AUMCinf/AUCinf – TI

/2, where TI represents infusion duration and AUMC<sub>inf</sub> is the area under the moment curve from the time of first

dosing extrapolated to infinity.

AUC<sub>0-12 wk</sub>/AUC<sub>inf</sub> calculated as AUC<sub>0-12 wk</sub>/AUC<sub>inf</sub>

AUC%extrap Percent of AUC extrapolated to infinity in AUCinf

Following administration, C<sub>max</sub>. t<sub>max</sub>, CLST and TLST will be obtained directly from the experimental observations. If multiple maxima occur at equal concentrations after an infusion, the first temporal value will be used.

AUC<sub>0-14 day</sub>, AUC<sub>0-12 wk</sub> and AUC<sub>inf</sub> will be estimated using the linear trapezoidal rule.

Values of AUC<sub>0-14 day</sub> and  $C_{max}$  associated with Dose 1 Infusion 2 will be listed but excluded from descriptive statistics and statistical analysis if the time of the last concentration following Dose 1 Infusion 1 is outside  $\pm$  2 day window around Day 15.


Values of AUC<sub>0-12 wk</sub> will be listed but excluded from descriptive statistics and statistical analysis if the time of the last concentration following Dose 1 Infusion 2 is outside  $\pm$  2 week window around Week 12.

The terminal half-life,  $t_{1/2}$ , where determined, will be calculated as  $ln(2)/\lambda_z$ . The number of data points included in the regression will be determined by visual inspection, but a minimum of three data points in the terminal phase, excluding  $C_{max}$ , will be required to estimate  $\lambda_z$ .  $\lambda_z$  values (and consequently  $t_{1/2}$  and  $AUC_{inf}$  values) will be considered unreliable estimates if the time period over which an individual  $\lambda_z$  was required is less than twice the resultant  $t_{1/2}$  or the adjusted coefficient of determination 'Rsq' is less than or equal to 0.8. Additional exclusions of PK parameters, if any, will be described in the CSR.

# 5.3 EFFICACY

#### ACR20/50/70

The ACR composite score evaluates clinical improvement relative to an initial assessment for clinical trials in subjects with RA.

The ACR20 response is defined as at least 20% improvement compared to baseline for both swollen and tender joint counts (66/68 joint counts), as well as for at least 3 out of the following 5 additional parameters:

- Subject's Global Health Assessment
- Investigator's Global Health Assessment
- Subject's assessment of pain
- Health Assessment Questionnaire Disability Index (HAQ-DI)
- C-Reactive Protein (CRP)

ACR50 and ACR70 are defined in a similar fashion to ACR20 but require at least 50 and 70 percent improvement respectively. Method for handling missing data is described in the appendice 2.

#### DAS28-CRP

The DAS28-CRP is a composite measure of disease activity in RA. It is a continuous measure based on 28 DAS joints from the ACR, the Subject's Global Health Assessment score, and CRP, as follows:

DAS28-CRP =  $0.56*(TJC28)^{0.5} + 0.28*(SJC28)^{0.5} + 0.36*ln(CRP+1) + 0.014*SGH + 0.96$ 

where TJC28 is the tender joint count of the 28 joints in the DAS, SJC28 is the swollen joint count of the 28 joints in the DAS, CRP is in mg/L, and SGH is the Subject's Global Health Assessment in 0 to 100 scale.

If the CRP is at a non-detectable level, then replace it with the minimum detectable level.




# **DAS28-CRP Remission**

A subject will be considered to have achieved DAS28-CRP remission if the subject has a DAS28-CRP score less than 2.6.

# Health Assessment Questionnaire – Disability Index (HAQ-DI)

The HAQ-DI score is defined as the average of the scores from eight sub-domains (dressing / grooming, arising, eating, walking, hygiene, reach, grip, and activities). The detailed score algorithm is described in Appendix 4.

# **Hybrid ACR Response**

Hybrid ACR response is a continuous score of the mean improvement in the core set measures combining the ACR20, ACR50, and ACR70 response rates.

The hybrid ACR can be calculated when all 7 components are available following the table below (American College of Rheumatology Committee to Reevaluate Improvement Criteria, 2007):

| | Mean % change in all 7 core set measures | | | |
|---|---|---|---|---|
| ACR Status | <20 | >=20, <50 | >=50, <70 | >=70 |
| Not ACR20 | Mean % change | 19.99 | 19.99 | 19.99 |
| ACR20 but not ACR50 | 20 | Mean % change | 49.99 | 49.99 |
| ACR50 but not ACR70 | 50 | 50 | Mean %<br>change | 69.99 |
| ACR70 | 70 | 70 | 70 | Mean %<br>change |

If a core set measure worsens by > 100%, the percentage change will be limited to 100%.

# Swollen Joint Count

The swollen joint count will be the number of joints that are assessed as swollen among the 66 joints specified in Section 17.3 of the protocol and the corresponding Joint Assessment CRF page. Method for handling missing joint assessments (including those due to artificial/fused joint or intra-articular corticosteroid injection) is defined in Appendix 3.

#### **Tender Joint Count**

The tender joint count will be the number of joints that are assessed as Pain/Tenderness among the 68 joints specified in Section 17.3 of the protocol and the corresponding Joint Assessment CRF page. Method for handling missing joint assessments (including those due to artificial/fused joint or intra-articular corticosteroid injection) is defined in Appendix 3.


# 5.4 SAFETY

# **Adverse Event of Interest (AEOI)**

An AEOI is defined as a noteworthy TEAE for a particular product or class of products that a sponsor may wish to monitor carefully. It could be serious or non-serious, and could include events that might be potential precursors or prodromes for more serious medical conditions in susceptible individuals (Council for International Organizations of Medical Sciences [CIOMS] VI, 2005). The AEOIs for this study will include:

- infusion reactions including hypersensitivity,
- cardiac disorders,
- serious infections,
- progressive multifocal leukoencephalopathy,
- hematological reactions,
- hepatitis B reaction,
- opportunistic infections
- hypogammaglobulinemia.
- severe mucocutaneous reactions.
- gastrointestinal perforation

Events of interest were identified using the latest versions of pre-specified Standardised MeDRA query (SMQ) where available. If no SMQ is available for use as a search tool for a given EOI (eg. Infusion reactions), a customized search strategy developed at Amgen or medical review will be used where SMQ is not available. Appendix 5 provides the search strategy used to retrieve the events of interest. The preferred terms used in the searches are stored in a central PRA server location for analyses.

# Exposure Adjusted Incidence Rate (EAIR) for Adverse Events and Adverse Event of Interest

The exposure adjusted incidence rate is defined as the number of subjects with a particular AE divided by the total exposure-time among subjects in the respective treatment group at risk of an initial occurrence of the event. Specifically,

Exposure Adjusted Incidence Rate = 
$$\frac{n}{T} = \frac{n}{\sum ti}$$
,

where n is the number of subjects with events, ti is a subject's exposure time under a given unit and T is the total exposure time under a given time unit of the subjects in the group. If a subject has multiple events, the ti is the time from the first dose date of the respective treatment to the onset of the first event. For those subjects who crossed over from one IP treatment during the 1<sup>st</sup> dose to another IP treatment during the 2<sup>nd</sup> dose, the exposure time following each of the doses will be counted in the respective treatment




group. For a subject with no event, the *ti* is set to the total exposure time duration of IP exposure (as defined in Section 5.1) for that subject.

# **Subject Incidence Rate**

For adverse event summaries, subject incidence rate for a given event is defined as the number of subjects with at least 1 reported occurrence of the event divided by the number of subjects that received the given treatment or total subjects for the total column. For subjects with multiple occurrences of the same event, the event will only be counted once per subject.

#### **Treatment-emergent Adverse Event**

A treatment-emergent AE (TEAE) is defined as an AE that begins or increases in severity or frequency at or after the first study IP administration through EOS. If the AE starts on the same day as the first dose of IP, then the flag indicating whether the AE started prior to the first dose on the adverse event CRF page will be used.

#### 5.5 PHARMACODYNAMICS

#### Complete depletion of CD19+ cell count

Complete depletion of CD19+ cell count at any post-dose time is defined as CD19+ cell counts < 20 cell/uL (0.02 x10^9 cell/L). Subjects with missing CD19+ cell count at baseline or subjects with CD19+ cell count < 20 cell/uL at baseline will be excluded from the derivation of complete depletion of CD19+ cell count.

#### **Duration of CD19+ B-cell complete depletion**

This variable will be defined only for subjects who had a CD19+ B-cell complete depletion for at least one post-dose time. It is defined as time from the first incidence of complete depletion of CD19+ cell count to when CD 19+ cell count first increases to >=20 cell/uL. Subjects whose CD 19+ cell count doesn't increase to >=20 cell/uL will be censored at the last CD19 assessment date.

# 6. ANALYSIS SETS

The primary statistical analysis for the PK endpoints will be based on the PK parameter analysis set. Sensitivity analysis for the PK endpoints will be based on the per-protocol (PP) PK parameter analysis set. The primary statistical analysis for the PD endpoint and efficacy endpoints will be performed using the full analysis set (FAS). The Per-protocol analysis set will be used for sensitivity analyses of the key efficacy endpoints. The analysis of safety endpoints will be based on the safety analysis set. The immunogenicity analysis will be based on anti-drug antibody analysis set.

#### 6.1 FULL ANALYSIS SET

The FAS includes all subjects randomized in the study, with treatment assignment based on treatment the subject is randomized to (regardless of actual treatment received).




# 6.2 PER-PROTOCOL ANALYSIS SET

The per-protocol (PP) analysis set includes all randomized subjects who have had two full infusions for the 1<sup>st</sup> dose (drug compliance of 90%-110%), have completed the week 24 disease assessment (complete DAS28-CRP assessment in the week 24 window of day 106-210 and before the 1st infusion of the 2nd dose), and did not experience a protocol deviation up to week 24 that affects their evaluation for the secondary objectives of the study to assess clinical efficacy. The protocol deviations that affect evaluation of the secondary objectives will be determined based on a blinded data review prior to database lock. Analyses for the per-protocol analysis set will be based on actual treatment received.

# 6.3 SAFETY ANALYSIS SET

The safety analysis set includes all randomized subjects who received at least 1 infusion of IP, with treatment assignment based on actual treatment received.

# 6.4 PHARMACOKINETIC CONCENTRATION ANALYSIS SET

The PK concentration analysis set is defined as the subset of subjects in the safety analysis set who received the full protocol-specified dose on Day 1 and had at least one evaluable serum concentration (including results below the quantifiable limit) of ABP 798 or rituximab. Pharmacokinetic concentration data from subjects will be analyzed according to the actual treatment received. Subjects to be excluded from the PK concentration analysis set will be determined based on a blinded data review prior to database lock.

#### 6.5 PHARMACOKINETIC PARAMETER ANALYSIS SET

The PK parameter analysis set is defined as the subset of subjects in the safety analysis set who received the full protocol-specified dose on Day 1 and had an evaluable ABP 798 or rituximab serum concentration time profile. The PK parameter analysis set will be used for the primary statistical analysis of PK endpoints. Pharmacokinetic parameter data from subjects will be analyzed according to the actual treatment received. Subjects to be excluded from the PK parameter analysis set will be determined based on a blinded data review prior to database lock.

# 6.6 PER-PROTOCOL PHARMACOKINETIC PARAMETER ANALYSIS SET

The per-protocol PK parameter analysis set consists of a subset of subjects in the PK parameter analysis set who do not experience an important protocol deviation that affects their PK evaluation. It will be analyzed according to actual treatment received. The important protocol deviations that affect evaluation of PK endpoints will be determined based on a blinded data review prior to database lock.




# 6.7 ANTI-DRUG ANTIBODY ANALYSIS SET

Anti-drug antibody analysis set is defined as the subset of subjects in the safety analysis set who had at least 1 evaluable antibody test. Immunogenicity data from subjects will be analyzed according to the actual treatment received.

# 7. INTERIM ANALYSES

No interim analyses are planned for this study.

A Data Monitoring Committee (DMC) external to Amgen and PRA will be formed with members consisting of individuals chosen for their expertise in inflammatory disorders. Members of the DMC will include, at a minimum, physicians external to Amgen and PRA, and appropriate statistical representation external to Amgen and PRA. The primary role of this independent DMC will be to monitor safety data.

The DMC will review unblinded safety data at regular intervals, as outlined in the DMC charter (approximately twice yearly; the start date will depend on subject accrual rates). The DMC will also review an initial safety analysis after the first 18 subjects have received the first dose.

In addition, the DMC will communicate major safety concerns and recommendations regarding study modification or termination to Amgen management at any time during the conduct of the study.

Details regarding the DMC will be provided in the DMC charter and DMC analysis plan.

# 8. DATA REVIEW

#### 8.1 DATA HANDLING AND TRANSFER

Data will be entered and exported as SAS® version 9.4 or higher datasets. Converted datasets will be created using SAS® and following standard Clinical Data Interchange Standards Consortium Standard Data Tabulation Model (CDISC SDTM, version 1.3, Implementation Guide version v3.1.3) conventions. Analysis datasets will be created using SAS® and following CDISC Analysis Data Model (ADaM, version 2.1, Implementation Guide 1.0) standards.

Medical history and AEs will be coded using the current version of MedDRA at the time of the analysis to assign a system organ class (SOC) and preferred term (PT) to each event. Adverse events and abnormal laboratory results considered as AEs are assigned a toxicity grade according to National Cancer Institute (NCI-US) Common Terminology Criteria for Adverse Events (CTCAE). Prior and concomitant medications will be coded using the current version of the World Health Organization Drug Dictionary (WHO-DD) at the time of the analysis.

Additional details can be found in the PRA Data Management Plan for this study.




# 8.2 DATA SCREENING

Beyond the data screening built into the PRA Data Management Plan, the PRA programming of analysis datasets and tables, figures and listings (TFLs) provides additional data screening as described below.

Review of a post-freeze dry run of TFLs allows for further data screening prior to final database lock for the entire study. This dry run will be discussed with the sponsor in data review meetings to identify any final data issues and seek corrections prior to the final database lock for the entire study. The PRA statistician and the sponsor must approve database lock.

# 9. STATISTICAL METHODS

All statistical analyses will be performed using SAS® (Version 9.4 or higher).

The final analysis will be performed after all subjects have completed or have had the opportunity to complete the week 48/EOS assessment.

Unless otherwise specified, descriptive data summaries will be tabulated by treatment for all endpoints. Categorical data will be summarized using number of subjects (n), frequency and percentages of subjects falling into each category, with the denominator for percentages being the number of subjects in the study population for each treatment group, unless otherwise noted. Percentages will be rounded to one decimal place. Confidence intervals will be provided where specified.

All continuous variables will be summarized using mean, standard deviation, median, minimum, maximum, 25th percentile (Q1), 75th percentile (Q3), and number of subjects with observations. The mean, median, Q1, and Q3 will be presented to one decimal place greater than the original data, standard deviation will be to two decimal places greater than the original data, and the minimum and maximum will have the same number of decimal places as the original data. Confience intervals will be provided where specified.

For any of the summaries that are to be done by visit, the derived analytical study visit as defined in section 5.1 will be used for analysis unless otherwise noted.

# 9.1 SUBJECT DISPOSITION

The following information will be summarized for subject disposition and accountability:

- Number of subjects randomized will be tabulated by region, country and center based on the FAS.
- Number of subjects randomized will be tabulated by stratification factors based on the FAS.
- Subject disposition (including number randomized, treated with ABP 798/rituximab (US)/rituximab (EU), completed treatment, discontinued treatment with reason of discontinuation, completed study, and discontinued study with reason of discontinuation) using each of the analysis sets defined in Section 6.


• Summaries of analysis sets with reason for exclusion for all screened subjects.

• Randomization list of subjects and their actual versus randomized treatment group for all randomized subjects.

# 9.2 PROTOCOL DEVIATIONS

Protocol deviation (PD) data will be entered into the Clinical Trials Management System (CTMS). The study team will conduct on-going reviews of the PD data from CTMS. The per-protocol analysis set and per protocol PK parameter analysis set must be finalized at the post-freeze data review meeting (or earlier), prior to the database lock.

Based on the PD data entered into CTMS, a summary of important PDs will be tabulated using number and percentage of subjects with important PD by deviation type and randomized treatment arm. A listing of subjects with important PDs will be provided (with a flag indicating whether the deviation leads to exclusion from the per-protocol and per-protocol pharmacokinetic analysis sets). A summary table and listing of eligibility criteria deviations will also be tabulated showing the violations of the inclusion/exclusion criteria for each subject.

# 9.3 TREATMENTS

# 9.3.1 Extent of IP Exposure

For the IP (ABP 798, rituximab (US) or rituximab (EU)), summary statistics will be provided for the total number of doses administered, total dose received, total duration of IP exposure, number of subjects with four full infusions and number of subjects with at least one partial infusion (including missed infusion), number of subjects with at least one infusion delay, number of subjects with at least one infusion missed, and number of subjects with at least one infusion interruption by treatment group. An IP administration summary will also be provided by the reported visit for each dosing/infusion instance, with summaries of the number of subjects receiving a full or partial infusion, infusion delay, infusion missed and infusion interruption as well as reasons, and reasons for ending IP by treatment group. The percentages for the IP administration summary will be based on the number of subjects with the given visit. The analysis will be performed using the safety analysis set according to the actual treatment received.

A subject listing of each administered lot number(s) for IP and a listing of unique manufacturing lot numbers used in the study will be provided.

# 9.3.2 Prior and Concomitant Medications

Prior and concomitant medications will be coded by WHO-DD and will be summarized by preferred name and treatment group. The prior medications and concomitant medications will be summarized by treatment groups. The analysis will be performed using the safety analysis set according to the actual treatment received.

The number and percentage of subjects using each medication will be displayed by treatment arm. Subjects taking more than one medication in the same preferred name will be counted once for the number of subjects taking that preferred name.


# 9.4 DEMOGRAPHIC AND BASELINE CHARACTERISTICS

The following demographics and baseline characteristics will be summarized by treatment for each of the analysis sets defined in Section 6.

- age (in years, at time of signing informed consent) and age category ( $<65 \text{ vs} \ge 65$ ),
- race,
- sex,
- ethnicity,
- height,
- weight,
- body mass index (BMI),
- BSA,
- geographic region (North America, Eastern Europe, and Western Europe),
- Number of prior biologic use for RA (1 vs. >1),
- Number of prior biologic use for RA (1, 2, 3, etc.),
- seropositivity (RF-positive and/or CCP-positive vs. RF-negative and CCPnegative),
- Duration of RA (in years) and duration of RA category ( $<5, \ge 5$  years),
- DAS28-CRP,
- swollen joint count(66 and 28 counts)
- tender joint count, (68 and 28 counts)
- subject's global health assessment,
- investigator's global health assessment,
- subject's assessment of disease-related pain,
- HAQ-DI,
- CRP,
- use of oral corticosteroid at baseline (Yes/No),
- use of non-steroidal anti-inflammatory drug (NSAID) at baseline (Yes/No),
- baseline methotrexate dose.

Medical conditions at screening and the status of the medical condition at randomization (continuing versus resolved) will be summarized by SOC and PT and tabulated by treatment groups ABP 798/ABP 798, rituximab (US)/ABP 798, rituximab


(EU)/rituximab (EU) and total. The analysis will be performed using the safety analysis set according to the actual treatment received.

# 9.5 PHARMACOKINETIC ANALYSES

#### 9.5.1 Pharmacokinetic Concentrations

Serum rituximab and ABP 798 concentrations will be summarized descriptively by treatment and nominal sampling time point for the PK concentration analysis set. The following descriptive statistics will be calculated at each of the sampling times: arithmetic mean (mean), coefficient of variation (CV), SD, Q1, Q3, Geometric mean, Geometric CV, minimum, median, maximum and the number of measurements. For calculation of summary concentrations, values below the quantifiable limit (BOL) will be set to zero.

In the event that a subject does not receive the full protocol-specified infusion, subsequent PK samples may be considered not evaluable and excluded from the descriptive statistics and mean concentration-time profiles. In addition, if samples are collected with a substantial deviation from nominal time that impacts the presentation of PK data, they will be excluded from the PK concentration vs nominal time profile. The samples excluded from the PK concentration analysis will be determined based on a blinded data review prior to unblinding for the final analysis.

Individual and mean (±SD) serum concentration-time profiles of rituximab and ABP 798 will be presented graphically using nominal time by treatment on a semi-logarithmic and a linear scale.

# 9.5.2 Pharmacokinetic Parameters

PK parameters for ABP 798 and rituximab will be estimated using noncompartmental analysis methods with Phoenix WinNonlin® Version 6.4 or higher (Pharsight Corp., St. Louis, MO).

In the event that a subject does not receive the full protocol-specified infusion, subsequent PK samples may be considered not evaluable and thus certain PK parameters may not be reportable. In addition, if the full protocol-specified dose was given but there was a long dose interruption or unusually long infusion duration that was deemed to impact PK, the PK profile may be considered not evaluable. The subject exclusion from the PK parameter analysis set will be determined based on a blinded data review prior to unblinding for the final analysis. Any such exclusion will be clearly listed in the CSR along with justification for exclusion.

Pharmacokinetic parameters will be listed by subject and summarized descriptively by treatment for the PK parameter analysis set. The following descriptive statistics will be provided: n, arithmetic mean, SD, Q1, Q3, minimum, median and maximum. Only n, median, Q1, Q3, minimum and maximum will be reported for t<sub>max</sub>. In addition, geometric mean, and geometric CV will be calculated for AUC<sub>inf</sub>, AUC<sub>0-14 day</sub>, AUC<sub>0-12 wk</sub>, C<sub>max</sub>, CLST2, t<sub>1/2</sub>, \(\lambda\zeright\), CL, MRT, AUC%extrap and AUC<sub>last</sub>/AUC<sub>inf.</sub>

The serum PK parameters will be estimated from the individual concentration data for all subjects in the PK parameter analysis set. In estimating the PK parameters, BOL values at

Statistical Analysis Plan Sponsor: Amgen Inc.


the beginning of the profile will be set to zero. BQL values that occur after the first quantifiable point will be considered missing. Actual sampling times will be used in all computations.

#### PRIMARY STATISTICAL ANALYSIS

The PK similarity will be demonstrated by comparing the 90% CI for the GMR of test (ABP 798)-to-reference (US-licensed rituximab or EU-authorized rituximab) and rituximab [US] to rituximab [EU] for AUC<sub>inf</sub> and for C<sub>max</sub> following the second infusion of the first dose with the bounds of 0.8 to 1.25. Point estimates and CIs for the GMR will be estimated from an analysis of covariance model using the PK parameter analysis set. For AUC<sub>inf</sub> and C<sub>max</sub> after second infusion of the first dose, the point estimates and 90% CIs for the GMR for will be estimated using an analysis of covariance model adjusted for weight and geographic region. A sample SAS code for PROC MIXED is displayed below:



The geometric least square means for each treatment will be presented. The ratios of the geometric means for the comparison of the test treatment to the reference treatment will be obtained by exponentiating the difference of the means on the natural log scale. The CIs will be obtained by exponentiating the CI for the difference between the means on the log scale. Plots of the ratio of geometric means and 90% CI will be displayed. Additionally, the similarity between PK endpoints of rituximab (US) and rituximab (EU) will be evaluated as well. The GMRs and 90% CIs will be generated for other PK endpoints: AUC<sub>0-14 day</sub>, AUC<sub>0-12 wk</sub>, and C<sub>max</sub> after the first infusion of the first dose by using the same methods as stated above.

#### SENSITIVITY ANALYSES

A sensitivity analysis of all PK parameters will be analyzed similarly to the primary statistical analysis using the PP PK parameter analysis set.

In addition, the following sensitivity analyses will be performed on the PK parameter analysis set:

- The point estimates and CIs for the GMR will be estimated using a model similar to the primary statistical analysis model but excluding all covariates.
- The point estimates and CIs for the GMR will be estimated using the primary statistical analysis model for the subgroups of subjects with negative binding ADA status and negative neutralizing ADA status during first dose period.


# 9.6 PHARMACODYNAMICS ANALYSES

All pharmacodynamics analyses will be performed using the FAS according to randomized treatment.

#### 9.6.1 **CD19**

The pharmacodynamics similarity will be evaluated descriptively for the difference in percent of subjects with complete CD19+ cell depletion between test (ABP 798) and reference (US-licensed rituximab or EU-authorized rituximab) from day 1 to day 3. Subjects with baseline value less than 20 cell/uL or missing will not be evaluable for CD19+ depletion analyses. The point estimate, the 90% CI and the 95% CI will be provided for rate difference and will be estimated using a generalized linear model (specifically, a log-binomial regression model) with stratification factors as covariates. A sample SAS code for PROC GENMOD is displayed below:



Note: The contrasts in the estimate statement may need to be changed depending on the order of the treatments.

Descriptive statistics for CD19+ counts as well as change from baseline will be provided at day 2 and day 3.

In addition, for duration of CD19 complete depletion, KM estimates and 90% CIs will be calculated by randomized treatment group for event time quartiles.

# 9.6.2 IgA, IgG and IgM

The total IgA, IgG and IgM levels as well as change from baseline will be summarized descriptively by treatment and visit.

# 9.7 EFFICACY ANALYSES

All efficacy analysis will be performed using the FAS based on subject's randomized treatment. Sensitivity analysis of DAS28 at week 24 will also be performed using the per-protocol analysis set based on the actual treatment the subject received.

Analyses will be performed for two different time periods:

1. From day 1 until week 24 (efficacy analysis visit weeks 8, 12 and 24), only including results prior to 1<sup>st</sup> infusion of 2<sup>nd</sup> dose. Subjects who had the 1<sup>st</sup> infusion of 2<sup>nd</sup> dose prior to week 24 will have their efficacy endpoints data censored at the timing of 1<sup>st</sup> infusion of 2<sup>nd</sup> dose. For example, if disease


assessment is done at day 1 of week 16 and 1<sup>st</sup> infusion of 2<sup>nd</sup> dose is done on the same day, then the disease assessment on day 1 of week 16 will be included in modeling, but any disease assessment after that day will not be included.

2. Day 1 through EOS (efficacy analysis visit weeks 8, 12, 24, 40 and 48). Analyses will be performed separately for all subjects and the subgroup of subjects who received the 1<sup>st</sup> infusion of the 2<sup>nd</sup> dose at week 24 (i.e., excluding early retreatment subjects as defined in section 5.1).

If PK similarity is established between rituximab (US) and rituximab (EU), the 2 arms will be combined into a single reference arm for the primary assessment of clinical equivalence of DAS28-CRP change from baseline at week 24 between ABP 798 and rituximab. The results for ABP 798 vs. rituximab (EU) and ABP 798 vs. rituximab (US) will be provided for descriptive purposes. If PK similarity is not established, the ABP 798 arm will be compared to each of the individual rituximab arms separately to establish clinical equivalence of ABP 798 to the individual reference arms.

The pooling of the reference arms for ACR20/50/70 and hybrid ACR analyses will be conducted similarly.

# 9.7.1 **DAS28-CRP**

#### PRIMARY STATISTICAL ANALYSIS

# DAS28-CRP at Week 24

The analyses will be performed on the FAS based on the day 1 through week 24 time period described above, with observed data. Subjects with missing baseline DAS28-CRP will not be included in the analysis since no change from baseline can be calculated. Analyses will assess the hypothesis that there are no clinically meaningful differences between ABP 798 and rituximab arms in DAS28-CRP change from baseline at week 24. This primary efficacy endpoint will be tested by comparing the 2-sided 90% CI of the change from baseline at week 24 of DAS28-CRP between ABP 798 and rituximab arms with an equivalence margin of (-0.6, 0.6).

To evaluate treatment differences across time points at which DAS28-CRP was assessed, repeated-measures analysis will be utilized for the day 1 through week 24 time period described above. Data from all assessed postbaseline time points will be included in the analysis. Besides stratification variables, baseline DAS28-CRP value, visit (week), treatment, and treatment-by-visit interaction will be included in the models, with visit as a categorical variable. The adjusted mean with 95% CI for each arm and 90% and 95% CIs for the mean difference will be constructed for mean difference of DAS28-CRP change from baseline between ABP 798 and rituximab arms at each time point.

The mixed model repeated measures analysis will be implemented using PROC MIXED in SAS. Because the time points at which measurements occur are not equally spaced (8, 12, and 24 weeks) and because measurements over time are expected to be correlated, with correlation coefficients being greater for time points that are closer together, a


spatial covariance structure denoted SP(POW) in SAS will be used. However, before implementing this structure, its appropriateness will be checked by choosing the smaller Akaike's information criterion when comparing the SP(POW) covariance structure with unstructured covariance structure. Example code for PROC MIXED with three treatment groups is displayed below:



Note: The contrasts in the Ismestimate statement may need to be changed depending on the order of the treatments. Only the individual arm comparison SAS code is presented.

# **DAS28-CRP at Other Time Points**

For time period from Day 1 to EOS, the treatment difference and its confidence intervals will be estimated using an ANCOVA model with baseline DAS28-CRP measurement and stratification factors as covariates at each visit window. A sample SAS code for ANCOVA model using PROC MIXED is displayed below:



Note: The contrasts in the estimate statement may need to be changed depending on the order of the treatments. Only the individual arm comparison SAS code is presented.

#### SENSITIVITY ANALYSES

To assess the robustness of the DAS28-CRP at week 24 results, the repeated measures analysis described above will be repeated using the PP analysis set based on the day 1 through week 24 time period described above. In addition, DAS28-CRP change from




baseline at week 24 will be analyzed using ANCOVA adjusting for stratification factors and baseline DAS28-CRP results.

A sensitivity analysis will also be done to explore the impact of the baseline covariates in section 9.4 on DAS28-CRP at week 24 in addition to the stratification factors. A stepwise model selection (with <0.25 p-value to enter the model and <0.1 to stay in the model) will be fit using PROC GLM and will be used to determine if any of the covariates have significant impact on the outcome variable. The final repeated measures model will be fit using PROC MIXED and will maintain treatment, the stratification factors, baseline DAS28-CRP, visit and visit by treatment regardless and the covariates identified by the stepwise model and the same covariance structure selected in the primary statistical analysis regardless. This additional exploration will be performed on the FAS based on the day 1 through week 24 time period described above.

Additional sensitivity analysis considering the drop-out and missing value will be described in the section 9.7.4.

In addition, for each subgroup (described in section 4.4) the DAS28-CRP at week 24 will also be examined in the subgroups. These additional explorations will be performed on the FAS based on the day 1 through week 24 time period described above by using the repeated measures analysis with the same covariance structure chosen in the primary statistical analysis. The 90% CI and 95% CIs of difference in mean change from baseline of DAS28-CRP will be displayed.

The DAS28-CRP change from baseline will be plotted by treatment and visit for the FAS with adjusted mean and 95% CI.

# 9.7.2 ACR 20/50/70

The analyses of ACR20/50/70 are descriptive. The RR of ACR20/50/70 at week 8, week 12 and week 24 (refers to the analysis visit) will be analyzed based on the day 1 through week 24 time period using a repeated measures analysis, where data are included as observed for both FAS and PP, unless otherwise specified. Besides stratification variables, visit week (as a categorical variable), treatment, and treatment-by-visit interaction will be included in the generalized estimating equation (GEE) model assuming a log link and an AR (1) correlation structure. Both 90% CI and 95% CI will be provided.

A sample SAS code for PROC GENMOD with the repeated statement is displayed below:





Statistical Analysis Plan Sponsor: Amgen Inc.


Note: The contrasts in the estimate statement may need to be changed depending on the order of the treatments. Only the individual arm comparison SAS code is presented.

The risk difference (RD) of ACR20 at week 8, week 12 and week 24 between ABP 798 and rituximab arms and corresponding 90% and 95% CIs will be displayed based on a GEE model similar to the above model with the link function changed to 'link=identity' and without the exponential transformation option under LSMESTIMATE and LSMEANS statement.

From Day 1 to EOS, the RR of ACR20/50/70 between ABP 798 and rituximab arms and their corresponding CIs will be estimated at each visit (weeks 8, 12, 24, 40 and 48) using generalized linear model (specifically, a log-binomial regression model) adjusted for the stratification factors as covariates with observed data. A sample SAS code for PROC GENMOD is displayed below:



Note: The contrasts in the estimate statement may need to be changed depending on the order of the treatments. Only the individual arm comparison SAS code is presented.

The RD of ACR20 between ABP and rituximab arms and their corresponding CIs will be obtained, based on a similar generalized linear model with link function changed to 'link=identity' and without the exponential transformation option under LSMESTIMATE and LSMEANS statements.

The adjusted percent of subjects achieving ACR20/50/70 will be plotted by treatment and week for the FAS accordingly.

# 9.7.3 Hybrid ACR

The analyses of hybrid ACR are descriptive. The mean difference of hybrid ACR score at week 8, week 12 and week 24 (refers to the analysis visit) will be analyzed using a repeated measures analysis described in section 9.7.1. From Day 1 to EOS, the mean difference and its confidence intervals will be estimated using an ANOVA model with stratification factors as covariates at each visit window. A similar sample SAS code for it is displayed in section 9.7.1.

Statistical Analysis Plan Sponsor: Amgen Inc.


# 9.7.4 Methods for Handling Dropouts and Missing Data for Efficacy

For ACR, the determination of ACR20/50/70 response will be based on the data available at each visit (refer to Appendix 2 for handling missing ACR individual components), taking into account prorated tenderness and swollenness of joints.

For the primary DAS28-CRP analysis, the primary repeated measures model will be fit to the observed data. The rate of missing DAS28-CRP at week 24 will be tabulated with reasons, such as missing baseline, incomplete week 24 assessment (missing up to 3 of 4 components), outside of the defined week 24 analysis time frame, missing week 24 component assessments (missing all 4 components), and discontinued from the study early prior to week 24 (day 210).

Tipping point analyses will be performed for the efficacy endpoints of DAS28-CRP change from baseline at week 24 based on ANCOVA model using FAS analysis set to explore the sensitivity of results to violations in assumptions about the missing data (i.e., to various missing not-at-random assumptions). Assumptions (tipping point) under which the 90% CI no longer rules out unacceptable differences in efficacy as determined by DAS28-CRP change from baseline at week 24 between ABP 798 and reference (Rituximab (US) and Rituximab (EU)) will be identified.

In this analysis, all the observed data will be included as non-missing, regardless of adherence to treatment or use of prohibited medication. The analysis will be performed using a general three-step approach:

- (1) Multiple imputation will be done using PROC MI to generate multiple (e.g., 10) imputed datasets by imputing missing data assuming monotone missing pattern and that subjects with missing data have, on average, worse or better efficacy compared to those who have values. The mean difference between the (unobserved) missing values and observed values (refer to as shift) can vary independently for the different treatment groups. For this analysis, the shifts for Rituximab(EU) and Rituximab(US) are assumed to be the same.
- (2) Each of these imputed datasets (which contains identical values of non-missing data but different values imputed for missing data) is analyzed using standard SAS procedure, e.g., PROC GLM, PROC GENMOD, etc.
- (3) Results from all imputed datasets are then combined together for overall inference using PROC MIANALYZE.

For DAS28-CRP change from baseline at week 24, seven equally spaced shifts (-0.9 to 0.9 by 0.3) for the DAS28-CRP change from baseline for subjects with missing data will be explored. A sample SAS code for given shifts is given as follows:


Statistical Analysis Plan Sponsor: Amgen Inc.




Note: Only the individual arm comparison SAS code is presented.

## 9.7.5 Multiplicity

No multiplicity adjustment will be done for efficacy endpoints.

## 9.7.6 Pooling of Sites

All sites will be pooled together for all analyses.

#### 9.8 SAFETY ANALYSES

All safety analyses will be performed on the Safety analysis set based on subject's actual treatment received. In general, summaries will be provided separately for (1) day 1 to 1st infusion of the 2nd dose of IP (exclusive) for subjects who received 2nd dose or to week 24 (day 175) or EOS (whichever is earlier) for subjects who didn't receive 2nd dose and (2) entire study, unless otherwise specified.

#### 9.8.1 Adverse Events

All reported AEs will be coded to the appropriate SOC and PT according to the most current version of MedDRA, and the severity of each AE will be graded by the investigator per CTCAE v4.03 criteria.

Only TEAE will be tabulated.

Subject incidence of the following AEs will be tabulated by treatment groups and by SOC, PT, and maximum severity grade per CTCAE v4.03:

• treatment-emergent AEs

Subject incidence of the following AEs will be tabulated by treatment groups and by SOC and PT:


treatment-emergent AEs

Subject incidence of the following AEs will be tabulated by preferred term in descending order of frequency in the ABP798 column:

- treatment-emergent AEs
- grade 3 or higher treatment-emergent AEs
- treatment-emergent AEs leading to discontinuation of IP/study
- treatment-emergent AEs leading to infusion delay/infusion not given
- treatment-emergent AEOIs

For treatment-emergent AEOIs, the point estimate and 95% CI for RD of the subject incidence between ABP and the reference product are provided.

Exposure adjusted subject incidence rate (EAIR) of the following AEs will be tabulated by preferred term in descending order of frequency in the ABP798 column for the entire study:

- treatment-emergent AEs
- treatment-emergent AEOIs

The point estimate and 95% CI for RR of the EAIR between ABP and the reference product are also provided.

AEs leading to discontinuation of IP/study are those with an action taken with Investigational Medicinal Product of "dose discontinued" or those with other action taken of "discontinued from study". If subjects have an AE for action taken with Investigational Medicinal Product of "dose delayed/not administered" checked, that AE leads to the infusion delay/infusion not given. If an AE leads to multiple actions taken with IP, only the last action will be captured in the eCRF.

Counting of AEs will be by subject, and subjects will be counted only once within each SOC or PT. For tables categorized by severity, subjects with multiple events within a particular SOC or preferred term will be counted under the category of their most severe event with that SOC or preferred term.

An overall summary table of treatment-emergent AEOIs will be displayed, providing the number and percent of subjects that are within each AEOI category. In addition, infusion reaction EOIs will also be summarized by PT and maximum CTCAE grade and also by infusion and PT.

A subject listing of AEs leading to discontinuation of IP/ study will be provided.

#### 9.8.2 Deaths and Serious Adverse Events

Subject incidence of the following will be tabulated by SOC, PT and maximum severity grade per CTCAT V4.03:

serious treatment-emergent AEs


Subject incidence of the following will be tabulated by preferred term in descending order of frequency of the ABP798 arm:

- serious treatment-emergent AEs
- treatment-emergent fatal AEs

A subject listing of SAEs and AEs with fatal outcome will be also provided.

## 9.8.3 Laboratory Data

Laboratory test results are reported in International System of Units (SI) units. Laboratory values and change from baseline will be summarized using descriptive statistics at each analysis visit by treatment. Shift tables of the worst on-study laboratory toxicity based on CTCAE v4.03 grading relative to baseline will be presented by treatment group. The shift tables will take into account all post-baseline (schedule and unscheduled) laboratory results for determination of worst on-study laboratory toxicity within the two summary timeframes listed previously. For labs with toxicity grading in two directions, for toxicity due to decreased value, the maximum grade is corresponding to the minimum post-baseline value. For toxicity due to increase value, the maximum grade is corresponding to the maximum post-baseline value. In addition, subject incidence tables and listings of grade  $\geq 3$  laboratory toxicities will be provided based on all post-baseline (scheduled and unscheduled) laboratory results for each of the two reporting periods. Standard ranges will be used for the laboratory analysis.

Lab assessments will be grouped for summary as follows:

- Hematology white blood cell parameters: white blood cell count and differential
- Hematology red blood cell parameters: hemoglobin, packed cell volume or hematocrit, red blood cell count, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration
- Hematology other parameters: platelets
- Serum chemistry hepatobiliary parameters: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase, gamma glutamyl transferase
- Serum chemistry general chemistry: sodium, potassium, albumin, total protein, non-fasting glucose
- Serum chemistry renal function tests: urea, creatinine

# 9.8.4 Vital Signs and Physical Examination

Observed and change from baseline in vital signs will be summarized by parameter and treatment. Descriptive statistics will be shown for baseline, each post-baseline time point up to EOS, and the change from baseline to each post-baseline time point.




## 9.8.5 Immunogenicity

The number and percentage of subjects developing binding and neutralizing ADA will be tabulated by treatment .

Pre-existing antibody incidence and developing antibody incidence will be summarized. Pre-existing antibody is defined as a positive antibody result at baseline (see Section 5.1 for definition of baseline). Developing antibody incidence is defined as a negative or no binding antibody result at baseline and a positive antibody result at a post-baseline time point. A transient antibody result is defined as a positive post-baseline result with a negative result at the subject's last time point tested within the study period.

In addition, the frequency and percent of subjects with positive binding or neutralizing ADA results will be tabulated by visit and treatment.

### 9.8.6 Methods for Handling Missing Data for Safety

Missing safety endpoints will not be imputed.

#### **Imputation for Partial or Missing Dates**

If dates are missing or incomplete for an AE (including deaths) or concomitant medication, the following algorithm will be used for imputation:

| | | Stop Date | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Complete: yyyymmdd | | Partial: yyyymm | | Partial: yyyy | | Missing |
| G D | | <1st | ≥1 <sup>st</sup> | <1st<br>dose<br>yyyym | ≥1 <sup>st</sup> dose | <1st<br>dose | ≥1 <sup>st</sup><br>dose | |
| Start Da | | dose | dose | m | yyyymm | уууу | уууу | |
| Partial : | = 1 <sup>st</sup><br>dose<br>yyyymm | 2 | 1 | n/a | 1 | n/a | 1 | 1 |
| yyyym<br>m | ≠ 1 <sup>st</sup> dose yyyymm | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Partial | = 1 <sup>st</sup><br>dose<br>yyyy | 2 | 1 | 3 | 1 | n/a | 1 | 1 |
| : <i>уууу</i> | ≠ 1 <sup>st</sup> dose yyyy | 3 | 3 | 3 | 3 | 3 | 3 | 3 |
| Missing | | 4 | 1 | 4 | 1 | 4 | 1 | 1 |

- **1** = Impute as the date of first dose
- **2** = Impute as the first of the month
- 3 =Impute as January 1 of the year
- **4** = Impute as January 1 of the stop year

Note: If the start date imputation leads to a start date that is after the stop date, then there is a data error and do not impute the start date.

Imputation rules for partial or missing stop dates:


1. Initial imputation

- a. For partial stop date "mmyyyy", impute the last of the month.
- b. For partial stop date "yyyy", impute December 31 of the year.
- c. For completely missing stop date, do not impute.
- 2. If the stop date imputation leads to a stop date that is after the death date, then impute the stop date as the death date.
- 3. If the stop date imputation leads to a stop date that is before the start date, then there is a data error and do not impute the stop date.

Imputation rules for partial or missing death dates:

- 1. If death year and month are available but day is missing:
  - a. If "mmyyyy" for last contact date = "mmyyyy" for death date, set death date to the day after the last contact date.
  - b. If "mmyyyy" for last contact date < "mmyyyy" for death date, set death date to the first day of the death month.
  - c. If "mmyyyy" for last contact date > "mmyyyy" for death date, data error and do not impute.
- 2. If both month and day are missing for death date or a death date is totally missing, set death date to the day after the last contact date.

The imputed dates will be used to assess whether AEs should be considered as treatment-emergent and if medications should be included in the safety summaries as prior or concomitant, however the original, partial dates will be included in data listings.

#### 9.9 EXPLORATORY ANALYSES

# 9.9.1 DAS28-CRP Individual Components

The DAS28-CRP individual components of swollen (28) and tender joint counts (28), subject's global health assessment, and CRP will be summarized as change from baseline descriptively by treatment and visit using the FAS as observed.

# 9.9.2 ACR Individual Components

The ACR individual components of swollen (66) and tender joint counts (68), subject's global health assessment, investigator's global assessment, subject's assessment of disease-related pain, HAQ-DI and CRP will be summarized descriptively by treatment and visit using the FAS as observed.

### 10. CHANGE FROM PROTOCOL SPECIFIED ANALYSIS

Druing the development of this document, pharmacokinetic concentration analysis set was defined in the SAP to better describe the analysis population criteria which will be the population set in the PK serum concentration TFLs. Additionally, the definition of per protocol and per protocol pharmacokinetic parameter analysis sets were modified to include "important protocol deviation" instead of "protocol deviation" to properly reflect the population included in this analysis set.


Furthemore, per protocol analysis set criteria also includes the condition of 2 full infusion of the first dose, meaning that the drug compliance of 90%-110% of the first dose, additionally to ensure this analysis set follows the protocol requirements.

#### 11. VALIDATION

The programming (including quality control) of the analysis datasets and TFLs will be conducted under PRA's standard processes PRS 050 and documented accordingly. The entire set of TFL will be checked for completeness and consistency prior to its delivery to the client by the lead statistician and a senior level statistician, or above, who is not a member of the project team.

The PRA validation process is repeated any time TFL are redelivered using different data. Execution of this validation process is documented through the study Table of Programs that is provided to the client at study conclusion.

#### 12. REFERENCES

Ke C, Wang J, Zhang C, Jiang Q, Snapinn S. On errors in stratified randomization. Statistics in Biopharmaceutical Research 2017; 9 (2): 225-33.

Volkmann ER, Agrawal H, Maranian P, Furst DE. Rituximab for rheumatoid arthritis: A meta-analysis and systematic review. Clin Med Insights: Therapeutics 2010:2 749-760. American College of Rheumatology Committee to Reevaluate Improvement Criteria, 2007, A 286 Proposed Revision to the ACR20: The Hybrid Measure of American College of Rheumatology Response, Arthritis Rheum., Mar 15;57(2):193-202




# APPENDIX 1 GLOSSARY OF ABBREVIATIONS

| | Glossary of Abbreviations: |
|---|---|
| ACR | American College of Rheumatology |
| ACR20 | 20% Improvement in ACR Core Set Measurements |
| ACR50 | 50% Improvement in ACR Core Set Measurements |
| ACR70 | 70% Improvement in ACR Core Set Measurements |
| ADA | Anti-drug Antibody |
| ADaM | Analysis Data Model |
| AEOI | Adverse Event of Interest |
| AE | Adverse Event |
| ALT | Alanine Aminotranferase |
| AST | Aspartate Aminotransferase |
| AUC | Area Under the Curve |
| BMI | Body Mass Index |
| BQL | Below Quantifiable Limit |
| ССР | Anti-cyclic Citrullinated Peptide |
| CDAI | Clinical Disease Activity Index |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CIOMS | Council for International Organizations of Medical Sciences |
| CL | clearance |
| C <sub>last</sub> | Last measurable Concentration |
| C <sub>max</sub> | Maximum Concentration |
| CRP | C-reactive Protein |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTMS | Clinical Trial Management System |
| CV | Coefficient of Variation |
| DAS | Disease Activity Score |
| DMARDs | Disease-modifying Anti-rheumatic Drugs |
| DMC | Data Monitoring Committee |
| eCRF | Electronic Case Report Form |
| EOI | End of Infusion |
| EOS | End of Study |
| EULAR | European League Against Rheumatism |
| FAS | Full Analysis Set |
| GEE | Generalized Estimating Equation |
| GH | General Health |



Sponsor: Amgen Inc.

Protocol No: 20130108

# Statistical Analysis Plan

10-December-2018/ Version 2.0

| GMR | Geometric Mean Ratio |
|---|---|
| HAQ-DI | Health Assessment Questionnaire Disability Index |
| IP | Investigational Product |
| IPD | Important protocol deviation |
| IXRS | Interactive Voice or Web Response System |
| IV | Intravenous |
| KM | Kaplan-meier |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRT | mean residence time |
| NCA | Noncompartmental techniques |
| NCI-US | National Cancer Institute |
| NSAID | Non-steroidal Anti-inflammatory Drug |
| PD | Pharmacodynamic |
| PD | Protocol Deviations |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PT | Preferred Term |
| Q1 | 25 <sup>th</sup> Percentile |
| Q3 | 75 <sup>th</sup> Percentile |
| RA | Rheumatoid Arthritis |
| RD | Risk Difference |
| RF | Rheumatoid Factor |
| RR | Risk Ratio |
| SAP | Statistical Analysis Plan |
| SAE | Serious Adverse Event |
| SDAI | Simplified Disease Activity Index score |
| SDTM | Standard Data Tabulation Model |
| SI | International System of Units |
| SJC28 | Swollen Joint Count (28 Joints) |
| SMQ | Standardised MedDRA Query |
| SOC | System Organ Class |
| t <sub>1/2</sub> | Terminal elimination half-life |
| TEAE | Treatment-emergent Adverse Event |
| TFL | Tables, Figures, and Listings |
| T <sub>max</sub> | Time to which the maximum serum concentration was observed |
| TJC28 | Tender Joint Count (28 Joints) |
| TNF | Tumor Necrosis Factor |




| VAS | Visual Analog Scale |
|--------|-------------------------------------------|
| WHO-DD | World Health Organization Drug Dictionary |
| λz | Terminal elimination rate constant |




# APPENDIX 2 METHOD FOR MISSING INDIVIDUAL COMPONENTS OF ACR CALCULATION

In the case of some ACR components are missing, the ACR composite scores will be based on the non-missing components. If a subject's non-missing components are not sufficient to identify ACR composite score, then that subject will be considered as missing ACR response. The corresponding algorithm is listed below (using ACR 20 as an example):

- If both Tender or Swollen Joint Counts are improved at least 20%, and
  - o If three or more of the other five ACR components are improved at least 20%, the subject is an ACR 20 responder;
  - o If three or more of the other five ACR components are not improved at least 20%, the subject is an ACR 20 non-responder;
  - o If none of the above, the ACR response for the subject cannot be determined due to missing data and is therefore coded as missing.
- If either swollen or tender joint counts is not improved at least 20%, the subject is an ACR non-responder
- If either swollen or tender joint counts is missing and the other improved at least 20%,

and

- o If three or more of the other five ACR components are not improved at least 20%, the subject is an ACR 20 non-responder;
- Otherwise, the ACR response for the subject cannot be determined due to missing data and is therefore coded as missing


# APPENDIX 3 METHOD FOR MISSING INDIVIDUAL JOINT ASSESSMENTS

A Pain/Tenderness or Swollen Joints may be coded as follows:

Joint 00 = None

**Codes:** 01 = Positive

08 = Permanently inevaluable because of replaced, fused joint

09 = Not evaluated because of intra-articular corticosteroid injection

77 = Not Done

The missing individual joint assessments due to artificial/fused joint, intra-articular corticosteroid injection or not done for other reason are imputed as the followings:

For Joint Codes = 08,

- At Screening: Code as missing at current visit only
- At Baseline: Exclude the joint from the total joint counts for baseline and all subsequent visits.
- Post-Baseline (If a joint is coded as 08 at a post-baseline visit but not at baseline): Code as "01" (failed) beginning with the current visit and all visits subsequent to the current visit.

For Joint Codes = 09,

- At Screening: Code as "01" (failed) at current visit only
- At Baseline: Code as "01" (failed) for baseline and all subsequent visits.
- <u>Post-Baseline</u>: Code as "01" (failed) beginning with the current visit and all visits subsequent to the current visit.

For Joint Codes = 77.

- <u>At Baseline</u>: Code as missing and exclude the joint from the total joint counts for baseline.
- Post-baseline: Code as missing and exclude the joint from the total joint counts for the current visit.

If there are joints being excluded after above imputation, the Tender or Swollen Joint Counts will be prorated based on the algorithm described below.




#### **Prorated Joint Counts**

If at least half but not all joints are evaluable (14 joints for the DAS28 joint counts, 34/33 for the 68/66 joint counts), then the observed prorated Tender or Swollen Joint Counts will be calculated. The prorated scores will be adjusted based upon the number of evaluable joints: the counted score will be multiplied by 28, 66, or 68 as applicable and divided by the number of joints evaluated. Otherwise, the Tender or Swollen Joint Counts is missing.

For example, if only 25 of the 28 DAS joints are assessed at a visit and 10 of those 25 are pain/tenderness and 8 of those 25 are swollen, the prorated joint counts are:

Tender Joint Counts: 10/25\*28 = 11.20 Swollen Joint Counts: 8/25\*28 = 8.96

That is, the values of 11.20 and 8.96 will be used in calculating the percent improvement, not the values of 10 and 8.



Statistical Analysis Plan Sponsor: Amgen Inc.


# APPENDIX 4 HAQ-DI SCORING ALGORTIHM

All language versions will use the following scoring system.

There are four possible responses for each sub-category item, or component, within a category:

0 =without ANY difficulty 2 = with MUCH difficulty

1 = with SOME difficulty 3 = UNABLE to do

- Step 1: Calculate the maximum score for each of the 8 categories (7 of the categories are listed in the table below. The eighth category "Activities" is not listed in the table due to lack of questions regarding use of aids or device). At least one question in each category needs to be answered to compute the maximum score.
- If an aid or device is used or help from another person is needed, set the score for the associated category to the maximum score between 2 and the score in step 1.

| Sub-domain | Aids or devices |
|---|---|
| Dressing&Grooming | Devices used for dressing (button hook, zipper pull, long-handled |
| | shoe horn, etc.) |
| Arising | Special or built up chair |
| Eating | Built up or special utensils |
| Walking | Cane, Walker, Crutches, Wheelchair |
| Hygiene | Raised toilet seat, Bathtub seat, Bathtub bar, Long-handled |
| | appliances in bathroom |
| Reach | Long-handled appliances for reach |
| Grip | Jar opener (for jars previously opened) |

If no more than 2 categories have missing scores, then the disability score is the mean of the non-missing category scores. Otherwise, the disability score is set to missing.




# APPENDIX 5 LIST OF EVENTS OF INTEREST AND THE ASSOCIATED SMQ AND EOI SEARCHING STRATEGIES

| | Category of EOI query | Search | Additional |
|---|---|---|---|
| | (SMQ, Amgen query, | Strategy | <b>Medical Review</b> |
| | or SOC) | | of the SMQ or |
| | | | SOC dataset for |
| Event of | | | confirmation of |
| Interest | | | the EOI |
| | Infusion reactions | Broad*- TEAE with start | |
| | (Amgen query) | date same as, or one day | |
| Infusion reactions | | after, IP administration date | No |
| including | Hypersensitivity (SMQ) | Broad- TEAE with start | 110 |
| Hypersensitivity | | date same as, or one day | |
| | | after, IP administration | |
| | | date | No |
| Cardiac disorders | Cardiac disorders (SOC) | | No |
| Serious infections | Infections and Infestations | | |
| | (SOC) | CTCAE grade >=3 or the | |
| Duo ano anizza | | serious TEAE | No |
| Progressive | D : 1:0 1 | | |
| multifocal | Progressive multifocal | | |
| leukoencephalopa | leukoencephalopathy | | |
| thy | (Amgen query) | Broad | Yes |
| Hematological | Hematopoietic cytopenia | | |
| reactions | (SMQ) | Broad | No |
| Hepatitis B | Hepatitis B Infection | | |
| reactivation | (Amgen query) | Broad | Yes |
| Opportunistic | Infections and infestations | | |
| infections | (SOC) | | Yes |
| | Immune mediated events | | |
| Hypogammaglob | associated with oncologic | | |
| ulinemia | immune therapies (Amgen | | |
| | query) | Broad | Yes |




| Severe | | | |
|---|---|---|---|
| mucocutaneous reactions | Severe cutaneous adverse reactions (SMQ) | CTCAE grade >=3 or the serious TEAE, Broad search | No |
| Gastrointestinal | Gastrointestinal | | |
| perforation | perforation(SMQ) | Narrow | No |

<sup>\*</sup>Broad search strategy includes both narrow scope terms and broad scope terms.




# APPENDIX 6 LIST OF POST-TEXT TABLES, FIGURES, LISTINGS, AND SUPPORTIVE SAS OUTPUT APPENDICES

| Table<br>Number | Table Title |
|---|---|
| 14.1 | Disposition and Analyzed Dataset Tables |
| Table 14.1.1 | Subject Analysis Sets by Treatment (All Screened Subjects) |
| Table 14-1.2.1. | Randomization by Region, Country and Center (Full Analysis Set) |
| Table 14-1.2.2. | Randomization by Stratification Factors (Full Analysis Set) |
| Table 14-1.3.1. | Subject Study Disposition by Treatment (Full Analysis Set) |
| Table 14- | |
| 1.3.2. | Subject Study Disposition by Treatment (Safety Analysis Set) |
| Table 14-1.3.3. | Subject Study Disposition by Treatment (Pharmacokinetic Concentration Analysis Set) |
| Table 14-1.3.4. | Subject Study Disposition by Treatment (Pharmacokinetic Parameter Analysis Set) |
| Table 14-1.3.5. | Subject Study Disposition by Treatment (Per Protocol Analysis Set) |
| Table 14-1.3.6. | Subject Study Disposition by Treatment (Per Protocol Pharmacokinetic Parameter Analysis Set) |
| Table 14-1.3.7. | Subject Study Disposition by Treatment (Anti-drug Antibody Analysis Set) |
| 14.2 | Demographic and Baseline Characteristics Data Tables |
| Table 14-2.1. | Demographic and Baseline Characteristics by Treatment (Full Analysis Set) |
| Table 14-2.2. | Demographic and Baseline Characteristics by Treatment (Safety Analysis Set) |
| Table 14-2.3. | Demographic and Baseline Characteristics by Treatment (Pharmacokinetic Concentration Analysis Set) |
| Table 14-2.4. | Demographic and Baseline Characteristics by Treatment (Pharmacokinetic Parameter Analysis Set) |
| Table 14-2.5. | Demographic and Baseline Characteristics by Treatment (Per<br>Protocol Analysis Set) |

Statistical Analysis Plan



Sponsor: Amgen Inc.

Protocol No: 20130108 10-December-2018/ Version 2.0 Demographic and Baseline Characteristics by Treatment (Per Table 14-2.6. Protocol Pharmacokinetic Parameter Analysis Set) Table 14-2.7. Demographic and Baseline Characteristics by Treatment (Anti-drug Antibody Analysis Set) Table 14-Resolved Medical Conditions at Randomization by System Organ Class, Preferred Term, and Treatment (Safety Analysis Set) 2.8.1. Table 14-Unresolved Medical Conditions at Randomization by System Organ 2.8.2. Class, Preferred Term, and Treatment (Safety Analysis Set) Table 14-2.9. Prior Medications by Preferred Name and Treatment (Safety Analysis Set) 14.3 **Measures of Treatment Compliance Data Tables** Table 14-3.1. Inclusion/Exclusion Criteria Protocol Deviations (Full Analysis Set) Table 14-3.2. Important Protocol Deviations (Full Analysis Set) Table 14-3.3. Concomitant Medications by Preferred Name and Treatment (Safety Analysis Set) 14.4 **Efficacy Data Tables** Repeated Measures Analysis of DAS28-CRP Change From Table 14-4.1.1. Baseline at Week 24 – Primary Analysis (Full Analysis Set) Analysis of DAS28-CRP Change From Baseline at Week 24 – Table 14-4.1.2. Sensitivity Analysis (Full Analysis Set) Repeated Measures Analysis of DAS28-CRP Change From Table 14-4.1.3.1. Baseline by Visit – Day 1 Through Week 24 (Full Analysis Set) Repeated Measures Analysis of DAS28-CRP Change From Table 14-4.1.3.2. Baseline by Visit – Day 1 Through Week 24 (Per Protocol Analysis Set) Table 14-4.1.4.1. Analysis of DAS28-CRP Change From Baseline by Visit – Day 1 Through End of Study (Full Analysis Set) Table 14-4.1.4.2. Analysis of DAS28-CRP Change From Baseline by Visit – Day 1 Through End of Study (Full Analysis Set – Subgroup who received the 1st infusion of the 2nd dose at week 24) Table 14-4.1.5. Summary for Reason of Missing DAS28-CRP Change from Baseline Results at Week 24 (Full Analysis Set) Table 14-4.1.6. Tipping Point Analysis Results for Mean Difference of DAS28-CRP Change From Baseline at Week 24 for ABP 798 vs Rituximab with 90% Confidence Interval (Full Analysis Set)

Statistical Analysis Plan



Sponsor: Amgen Inc.

Protocol No: 20130108 10-December-2018/ Version 2.0 Table 14-4.1.7. Repeated Measures Analysis with Additional Selective Covariates for DAS28-CRP Change From Baseline at Week 24 (Full Analysis Set) Repeated Measures Analysis of DAS28-CRP Change From Table 14-4.2.1. Baseline by Age Subgroup - Day 1 Through Week 24 (Full Analysis Set) Table 14-4.2.2. Repeated Measures Analysis of DAS28-CRP Change From Baseline by Race Subgroup – Day 1 Through Week 24 (Full Analysis Set) Table 14-4.2.3. Repeated Measures Analysis of DAS28-CRP Change From Baseline by Gender Subgroup – Day 1 Through Week 24 (Full Analysis Set) Table 14-4.2.5. Repeated Measures Analysis of DAS28-CRP Change From Baseline by Binding Anti-drug Antibodies Status Subgroup – Day 1 Through Week 24 (Full Analysis Set) Table 14-4.2.6. Repeated Measures Analysis of DAS28-CRP Change From Baseline by Neutralizing Anti-drug Antibodies Status Subgroup – Day 1 Through Week 24 (Full Analysis Set) Repeated Measures Analysis of DAS28-CRP Change From Table 14-4.2.7. Baseline by Baseline Oral Corticosteroid Use Subgroup – Day 1 Through Week 24 (Full Analysis Set) Repeated Measures Analysis of DAS28-CRP Change From Table 14-4.3.1. Baseline by Geographic Region Subgroup – Day 1 Through Week 24 (Full Analysis Set) Repeated Measures Analysis of DAS28-CRP Change From Table 14-4.3.2. Baseline by Seropositivity Subgroup – Day 1 Through Week 24 (Full Analysis Set) Table 14-4.3.3. Repeated Measures Analysis of DAS28-CRP Change From Baseline by Prior Biologics Use Subgroup – Day 1 Through Week 24 (Full Analysis Set) Table 14-4.5.1.1 Repeated Measures Analysis of ACR20 by Visit – Day 1 Through Week 24 (Full Analysis Set) Table 14-4.5.1.2 Repeated Measures Analysis of ACR20 by Visit – Day 1 Through Week 24 (Per Protocol Analysis Set) Table 14-4.5.2.1. Analysis of ACR20 by Visit – Day 1 Through End of Study (Full Analysis Set)



Statistical Analysis Plan Sponsor: Amgen Inc. Protocol No: 20130108 10-December-2018/ Version 2.0 Analysis of ACR20 by Visit – Day 1 Through End of Study (Full Table 14-4.5.2.2. Analysis Set – Subgroup who received the 1st infusion of the 2nd dose at week 24) Repeated Measures Analysis of Hybrid ACR by Visit – Day 1 Table 14-4.5.3.1 Through Week 24 (Full Analysis Set) Table 14-4.5.3.2 Repeated Measures Analysis of Hybrid ACR by Visit – Day 1 Through Week 24 (Per Protocol Analysis Set) Analysis of Hybrid ACR by Visit – Day 1 Through End of Study Table 14-4.5.3.3. (Full Analysis Set) Table 14-4.5.3.4. Analysis of Hybrid ACR by Visit – Day 1 Through End of Study (Full Analysis Set – Subgroup who received the 1st infusion of the 2nd dose at week 24) Table 14-4.6.1. Repeated Measures Analysis of ACR50 by Visit – Day 1 Through Week 24 (Full Analysis Set) Table 14-4.6.2.1. Analysis of ACR50 by Visit – Day 1 Through End of Study (Full Analysis Set) Analysis of ACR50 by Visit – Day 1 Through End of Study (Full Table 14-4.6.2.2. Analysis Set – Subgroup who received the 1st infusion of the 2nd dose at week 24) Repeated Measures Analysis of ACR70 by Visit – Day 1 Through Table 14-4.7.1. Week 24 (Full Analysis Set) Table 14-4.7.2.1. Analysis of ACR70 by Visit – Day 1 Through End of Study (Full Analysis Set) Table 14-4.7.2.2. Analysis of ACR70 by Visit – Day 1 Through End of Study (Full Analysis Set–Subgroup who received the 1st infusion of the 2nd dose at week 24) Table 14-4.8.1. Summary of Swollen Joint Counts by Visit (Full Analysis Set) Table 14-4.8.2. Summary of Tender Joint Counts by Visit (Full Analysis Set) Table 14-4.8.3. Summary of Subject's Global Health Assessment by Visit (Full Analysis Set) Summary of Investigator's Global Health Assessment by Visit Table 14-4.8.4. (Full Analysis Set) Summary of Subject's Assessment of Disease-related Pain by Table 14-4.8.5. Visit (Full Analysis Set) Summary of HAQ-DI Total Score by Visit (Full Analysis Set) Table 14-4.8.6.

Summary of CRP by Visit (Full Analysis Set)

Table 14-4.8.7.



| Table 14-4.8.8. | Summary of Swollen Joint Counts by Visit – DAS28-CRP<br>Component (Full Analysis Set) |
|---|---|
| Table 14-4.8.9. | Summary of Tender Joint Counts by Visit – DAS28-CRP<br>Component (Full Analysis Set) |
| Table 14-4.8.10. | Summary of Subject's Global Health Assessment by Visit – DAS28-CRP Component (Full Analysis Set) |
| Table 14-4.8.11. | Summary of CRP by Visit – DAS28-CRP Component (Full Analysis Set) |
| Table 14-4.10.1.1. | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline at Week 24 Comparing ABP 798 with Pooled Rituximab<br>(Full Analysis Set) |
| Table 14-4.10.1.2. | Analysis of DAS28-CRP Change From Baseline (ANCOVA) at Week 24 Comparing ABP 798 with Pooled Rituximab (Full Analysis Set) |
| Table 14-4.10.1.3.1. | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline Comparing ABP 798 with Pooled Rituximab by Visit –<br>Day 1 ThroughWeek 24 (Full Analysis Set) |
| Table 14-4.10.1.3.2. | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline Comparing ABP 798 with Pooled Rituximab by Visit –<br>Day 1 Through Week 24 (Per Protocol Analysis Set) |
| Table 14-4.10.1.4.1. | Analysis of DAS28-CRP Change From Baseline (ANCOVA)<br>Comparing ABP 798 with Pooled Rituximab by Visit – Day 1<br>Through End of Study (Full Analysis Set) |
| Table 14-4.10.1.4.2. | Analysis of DAS28-CRP Change From Baseline (ANCOVA)<br>Comparing ABP 798 with Pooled Rituximab by Visit – Day 1<br>Through End of Study (Per Protocol Set) |
| Table 14-4.10.1.6. | Tipping Point Analysis Results for Mean Difference of DAS28-CRP Change From Baseline at Week 24 for ABP 798 vs Pooled Rituximab with 90% Confidence Interval (Full Analysis Set) |
| Table 14-4.10.1.7. | Repeated Measures Analysis with Additional Selective Covariates for DAS28-CRP Change From Baseline at Week 24 Comparing ABP 798 with Pooled Rituximab (Full Analysis Set) |
| Table 14-4.10.5.1 | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline Comparing ABP 798 with Pooled Rituximab by Age<br>Subgroup - Day 1 Through Week 24 (Full Analysis Set) |
| Table 14-4.10.5.2 | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline Comparing ABP 798 with Pooled Rituximab by Race<br>Subgroup – Day 1 Through Week 24 (Full Analysis Set) |



Sponsor: Amgen Inc.

Protocol No: 20130108

Table 14-4.10.5.3 Repeated Measures Analysis of DAS28-CRP Change From

| Table 14-4.10.5.3 | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline Comparing ABP 798 with Pooled Rituximab by Gender<br>Subgroup – Day 1 Through Week 24 (Full Analysis Set) |
|---|---|
| Table 14-4.10.5.5 | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline Comparing ABP 798 with Pooled Rituximab by Binding<br>Anti-drug Antibodies Status Subgroup – Day 1 Through Week 24<br>(Full Analysis Set) |
| Table 14-4.10.5.6 | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline Comparing ABP 798 with Pooled Rituximab by<br>Neutralizing Anti-drug Antibodies Status Subgroup – Day 1<br>Through Week 24 (Full Analysis Set) |
| Table 14-4.10.5.7 | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline Comparing ABP 798 with Pooled Rituximab by<br>Baseline Oral Corticosteroid Use Subgroup – Day 1 Through<br>Week 24 (Full Analysis Set) |
| Table 14-4.10.6.1 | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline Comparing ABP 798 with Pooled Rituximab by<br>Geographic Region Subgroup – Day 1 Through Week 24 (Full<br>Analysis Set) |
| Table 14-4.10.6.2 | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline Comparing ABP 798 with Pooled Rituximab by<br>Seropositivity Subgroup – Day 1 Through Week 24 (Full Analysis<br>Set) |
| Table 14-4.10.6.3 | Repeated Measures Analysis of DAS28-CRP Change From<br>Baseline Comparing ABP 798 with Pooled Rituximab by Prior<br>Biologics Use Subgroup – Day 1 Through Week 24 (Full Analysis<br>Set) |
| Table 14-4.11.5.1.1 | Repeated Measures Analysis of ACR20 Comparing ABP 798 with Pooled Rituximab by Visit – Day 1 Through Week 24 (Full Analysis Set) |
| Table 14-<br>4.11.5.1.2 | Repeated Measures Analysis of ACR20 Comparing ABP 798 with Pooled Rituximab by Visit – Day 1 Through Week 24 (Per Protocol Analysis Set) |
| Table 14-4.12.1.1 | Repeated Measures Analysis of Hybrid ACR Comparing ABP 798 with Pooled Rituximab by Visit – Day 1 Through Week 24 (Full Analysis Set) |
| Table 14-4.12.1.2 | Repeated Measures Analysis of Hybrid ACR Comparing ABP 798 with Pooled Rituximab by Visit – Day 1 Through Week 24 (Per Protocol Analysis Set) |

Statistical Analysis Plan



Sponsor: Amgen Inc.

Protocol No: 20130108 10-December-2018/ Version 2.0 Repeated Measures Analysis of ACR 50 Comparing ABP 798 Table 14-4.13.1 with Pooled Rituximab by Visit – Day 1 Through Week 24 (Full Analysis Set) Repeated Measures Analysis of ACR 70 Comparing ABP 798 Table 14-4.14.1 with Pooled Rituximab by Visit – Day 1 Through Week 24 (Full Analysis Set) Figure 14-4.10. Mean DAS28-CRP Change from Baseline – Day 1 Through Week 24 (Full Analysis Set) Percent of Subjects Achieving ACR20 Response – Day 1 Through Figure 14-4.11.1. End of Study (Full Analysis Set) Percent of Subjects Achieving ACR50 Response – Day 1 Through Figure 14-4.11.2. End of Study (Full Analysis Set) Figure 14-4.11.3. Percent of Subjects Achieving ACR70 Response – Day 1 Through End of Study (Full Analysis Set) Figure 14-4.11.4. Mean Hybrid ACR – Day 1 Through End of Study (Full Analysis Set) Figure 14-4.11. ACR Response at Week 24 (Full Analysis Set) Mean DAS28-CRP Change from Baseline with Pooled Rituximab Figure 14-4.12. - Day 1 Through Week 24 (Full Analysis Set) Figure 14-4.13.1. Percent of Subjects Achieving ACR20 Response with Pooled Rituximab – Day 1 Through Week 24 (Full Analysis Set) Figure 14-4.13.2. Percent of Subjects Achieving ACR50 Response with Pooled Rituximab – Day 1 Through Week 24 (Full Analysis Set) Figure 14-4.13.3. Percent of Subjects Achieving ACR70 Response with Pooled Rituximab – Day 1 Through Week 24 (Full Analysis Set) Figure 14-4.13.4. Mean Hybrid ACR with Pooled Rituximab – Day 1 Through Week 24 (Full Analysis Set) 14.5 **Extent of Exposure Tables** Table 14-5.1. Investigational Product Exposure Summary by Treatment (Safety Analysis Set) Table 14-5.2. Investigational Product Administration by Visit and Treatment (Safety Analysis Set) 14.6 **Adverse Events Data Tables** Table 14-6.1.1. Overall Summary of Treatment-emergent Adverse Events by Treatment – Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set)



| Table 14-6.1.2. | Overall Summary of Treatment-emergent Adverse Events by<br>Treatment –Day 1 Through End of Study (Safety Analysis Set) |
|---|---|
| Table 14-6.2.1.1. | Treatment-emergent Adverse Events by System Organ Class,<br>Preferred Term, and Treatment – Day 1 Until 1st Infusion of 2nd<br>Dose (Safety Analysis Set) |
| Table 14-6.2.1.2. | Treatment-emergent Adverse Events by System Organ Class,<br>Preferred Term, and Treatment – Day 1 Through End of Study<br>(Safety Analysis Set) |
| Table 14-6.2.2.1. | Treatment-emergent Adverse Events by Preferred Term and Treatment – Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) |
| Table 14-6.2.2.2. | Treatment-emergent Adverse Events by Preferred Term and Treatment – Day 1 Through End of Study (Safety Analysis Set) |
| Table 14-6.2.2.3. | Treatment-emergent Adverse Events by Age Subgroup, Preferred<br>Term and Treatment – Day 1 Until 1st Infusion of 2nd Dose<br>(Safety Analysis Set) |
| Table 14-6.2.2.4. | Treatment-emergent Adverse Events by Age Subgroup, Preferred<br>Term and Treatment – Day 1 Through End of Study (Safety<br>Analysis Set) |
| Table 14-6.2.3.1. | Treatment-emergent Adverse Events by System Organ Class,<br>Preferred Term, Maximum CTCAE Grade, and Treatment – Day 1<br>Until 1st Infusion of 2nd Dose (Safety Analysis Set) |
| Table 14-6.2.3.2. | Treatment-emergent Adverse Events by System Organ Class,<br>Preferred Term, Maximum CTCAE Grade, and Treatment – Day 1<br>Through End of Study (Safety Analysis Set) |
| Table 14-6.2.4.1. | Grade ≥3 Treatment-emergent Adverse Events by Preferred Term and Treatment - Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) |
| Table 14-6.2.4.2. | Grade ≥3 Treatment-emergent Adverse Events by Preferred Term and Treatment – Day 1 Through End of Study (Safety Analysis Set) |
| Table 14-6.3.1.1. | Treatment-emergent Adverse Events Leading to Discontinuation of IP/Study by Preferred Term and Treatment – Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) |
| Table 14-6.3.1.2. | Treatment-emergent Adverse Events Leading to Discontinuation of IP/Study by Preferred Term and Treatment – Day 1 Through End of Study (Safety Analysis Set) |



Statistical Analysis Plan Sponsor: Amgen Inc. 10-December-2018/ Version 2.0 Protocol No: 20130108

| Table 14-6.3.1.3. | Treatment-emergent Adverse Events Leading to Infusion<br>Delay/Infusion Not Given by Preferred Term and Treatment –<br>Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) |
|---|---|
| Table 14-6.3.1.4. | Treatment-emergent Adverse Events Leading to Infusion<br>Delay/Infusion Not Given by Preferred Term and Treatment –<br>Day 1 Through End of Study (Safety Analysis Set) |
| Table 14-6.4.1.1. | Treatment-emergent Adverse Events with Fatal Outcome by Preferred Term and Treatment – Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) |
| Table 14-6.4.1.2. | Treatment-emergent Adverse Events with Fatal Outcome by Preferred Term and Treatment – Day 1 Through End of Study (Safety Analysis Set) |
| Table 14-6.4.2.1. | Serious Treatment-emergent Adverse Events by System Organ<br>Class, Preferred Term, Maximum CTCAE Grade and Treatment –<br>Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) |
| Table 14-6.4.2.2. | Serious Treatment-emergent Adverse Events by System Organ<br>Class, Preferred Term, Maximum CTCAE Grade and Treatment –<br>Day 1 Through End of Study (Safety Analysis Set) |
| Table 14-6.4.3.1. | Serious Treatment-emergent Adverse Events by Preferred Term<br>and Treatment – Day 1 Until 1st Infusion of 2nd Dose (Safety<br>Analysis Set) |
| Table 14-6.4.3.2. | Serious Treatment-emergent Adverse Events by Preferred Term<br>and Treatment – Day 1 Through End of Study (Safety Analysis<br>Set) |
| Table 14-6.5.1.1. | Overall Events of Interest Treatment-emergent Adverse Events by Treatment – Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) |
| Table 14-6.5.1.2. | Overall Events of Interest Treatment-emergent Adverse Events by Treatment – Day 1 Through End of Study (Safety Analysis Set) |
| Table 14-6.6.1.1.1. | Infusion Reactions Including Hypersensitivity Treatment-<br>emergent Adverse Events by Preferred Term – Day 1 Until 1st<br>Infusion of 2nd Dose (Safety Analysis Set) |
| Table 14-6.6.1.1.2. | Infusion Reactions Including Hypersensitivity Treatment-<br>emergent Adverse Events by Preferred Term – Day 1 Through<br>End of Study (Safety Analysis Set) |
| Table 14-6.6.1.2.1. | Cardiac Disorders Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Until 1st Infusion of 2nd Dose (Safety<br>Analysis Set) |



| 201301 | To December 2010/ Version 2.0 |
|---|---|
| Table 14-6.6.1.2.2. | Cardiac Disorders Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Through End of Study (Safety Analysis<br>Set) |
| Table 14-6.6.1.3.1. | Serious Infections Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Until 1st Infusion of 2nd Dose (Safety<br>Analysis Set) |
| Table 14-6.6.1.3.2. | Serious Infections Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Through End of Study (Safety Analysis<br>Set) |
| Table 14-<br>6.6.1.4.1. | Progressive Multifocal Leukoencephalopathy Treatment-emergent<br>Adverse Events by Preferred Term – Day 1 Until 1st Infusion of<br>2nd Dose (Safety Analysis Set) |
| Table 14-6.6.1.4.2. | Progressive Multifocal Leukoencephalopathy Treatment-emergent<br>Adverse Events by Preferred Term – Day 1 Through End of Study<br>(Safety Analysis Set) |
| Table 14-6.6.1.5.1. | Hematological Reactions Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Until 1st Infusion of 2nd Dose (Safety<br>Analysis Set) |
| Table 14-6.6.1.5.2. | Hematological Reactions Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Through End of Study (Safety Analysis<br>Set) |
| Table 14-6.6.1.6.1. | Hepatitis B Reactions Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Until 1st Infusion of 2nd Dose (Safety<br>Analysis Set) |
| Table 14-6.6.1.6.2. | Hepatitis B Reactions Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Through End of Study (Safety Analysis<br>Set) |
| Table 14-6.6.1.7.1. | Opportunistic infections Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Until 1st Infusion of 2nd Dose (Safety<br>Analysis Set) |
| Table 14-6.6.1.7.2. | Opportunistic infections Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Through End of Study (Safety Analysis<br>Set) |
| Table 14-6.6.1.8.1. | Hypogammaglobulinemia Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Until 1st Infusion of 2nd Dose (Safety<br>Analysis Set) |
| Table 14-6.6.1.8.2. | Hypogammaglobulinemia Treatment-emergent Adverse Events by<br>Preferred Term – Day 1 Through End of Study (Safety Analysis<br>Set) |



| Severe Mucocutaneous Reactions Treatment-emergent Adverse<br>Events by Preferred Term – Day 1 Until 1st Infusion of 2nd Dose<br>(Safety Analysis Set) |
|---|
| Severe Mucocutaneous Reactions Treatment-emergent Adverse<br>Events by Preferred Term – Day 1 Through End of Study (Safety<br>Analysis Set) |
| Gastrointestinal Perforation Treatment-emergent Adverse Events<br>by Preferred Term – Day 1 Until 1st Infusion of 2nd Dose (Safety<br>Analysis Set) |
| Gastrointestinal Perforation Treatment-emergent Adverse Events<br>by Preferred Term – Day 1 Through End of Study (Safety<br>Analysis Set) |
| Infusion Reactions Including Hypersensitivity Treatment-<br>emergent Adverse Events by Preferred Term, Maximum CTCAE<br>Grade, and Treatment – Day 1 Until 1st Infusion of 2nd Dose<br>(Safety Analysis Set) |
| Infusion Reactions Including Hypersensitivity Treatment-<br>emergent Adverse Events by Preferred Term, Maximum CTCAE,<br>and Treatment – Day 1 Through End of Study (Safety Analysis<br>Set) |
| Infusion Reactions Including Hypersensitivity Treatment-<br>emergent Adverse Events of Interest (EOI) by Infusion, Preferred<br>Term, and Treatment – Day 1 Through End of Study (Safety<br>Analysis Set) |
| Exposure Adjusted Incidence Rate for Treatment-emergent<br>Adverse Events by Preferred Term and Treatment - Day 1<br>Through End of Study (Safety Analysis Set) |
| Exposure Adjusted Incidence Rate for Treatment-emergent<br>Adverse Events of Interest by Treatment – Day 1 Through End of<br>Study (Safety Analysis Set) |
| Clinical Laboratory Tables |
| Hematology Results by Visit and Treatment – White Blood Cell<br>Parameters (Safety Analysis Set) |
| Hematology Results by Visit and Treatment – Red Blood Cell<br>Parameters (Safety Analysis Set) |
| Hematology Results by Visit and Treatment – Other Parameters (Safety Analysis Set) |

Statistical Analysis Plan



Sponsor: Amgen Inc.

Protocol No: 20130108 10-December-2018/ Version 2.0 Table 14-7.1.4.1. Shift Summary of Hematology Results by Maximum Postbaseline CTCAE Grade and Treatment – Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) Table 14-7.1.4.2. Shift Summary of Hematology Results by Maximum Postbaseline CTCAE Grade and Treatment – Day 1 Through Entire Study (Safety Analysis Set) Table 14-7.1.5.1. Incidence of Grade ≥3 Post-baseline Hematology Result by Treatment – Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) Table 14-7.1.5.2. Incidence of Grade ≥3 Post-baseline Hematology Result by Treatment – Day 1 Through End of Study (Safety Analysis Set) Serum Chemistry Results by Visit and Treatment – Hepatobiliary Table 14-7.2.1. Parameters (Safety Analysis Set) Table 14-7.2.2. Serum Chemistry Results by Visit and Treatment – General Chemistry (Safety Analysis Set) Table 14-7.2.3. Serum Chemistry Results by Visit and Treatment – Renal Function Tests (Safety Analysis Set) Shift Summary of Serum Chemistry Results by Maximum Post-Table 14-7.2.4.1. baseline CTCAE Grade and Treatment – Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) Table 14-7.2.4.2. Shift Summary of Serum Chemistry Results by Maximum Postbaseline CTCAE Grade and Treatment – Day 1 Through End of Study (Safety Analysis Set) Table 14-7.2.5.1. Incidence of Grade ≥3 Post-baseline Chemistry Result by Treatment – Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) Table 14-7.2.5.2. Incidence of Grade >3 Post-baseline Chemistry Result by Treatment – Day 1 Through End of Study (Safety Analysis Set) 14.8 **Other Safety Endpoints Data Tables** Vital Sign Results by Visit and Treatment (Safety Analysis Set) Table 14-8.1. 14.9 **Pharmacokinetics Data Table** Summary of ABP 798 Serum Concentrations (ug/mL) (PK Table 14-9.1.1. Concentration Analysis Set) Summary of Rituximab (US) Serum Concentrations (ug/mL) Table 14-9.1.2. (Through Week 24) and ABP 798 Serum Concentration (Week 26 Through End of Study) (PK Concentration Analysis Set) Table 14-9.1.3. Summary of Rituximab (EU) Serum Concentrations (ug/mL) (PK Concentration Analysis Set)



Statistical Analysis Plan Sponsor: Amgen Inc. Protocol No: 20130108 10-December-2018/ Version 2.0 Figure 14-9.4.1. Mean (+/-SD) Serum Concentrations Over Time by Treatment -Through Week 12 (PK Concentration Analysis Set) Figure 14-9.4.5. Boxplot of Trough ABP 798 Serum Concentration - Week 24 Through End of Study (PK Concentration Analysis Set) Individual ABP 798 Concentration (Linear)-Time Profiles for Figure 14-9.4.6.1. Subjects in the ABP798/ABP798 Arm - Through Week 12 (PK Concentration Analysis Set) Individual ABP 798 Concentration (Linear)-Time Profiles for Figure 14-9.4.7.1 Subjects in the Rituximab (US)/ABP798 Arm - Through Week 12 (PK Concentration Analysis Set) Figure 14-9.4.8.1 Individual Rituximab (EU) Concentration (Linear) - Time Profiles for Subjects in the Rituximab (EU)/Rituximab (EU) Arm -Through Week 12 (PK Concentration Analysis Set) Ratio of Geometric Means and 90% Confidence Intervals of PK Figure 14-9.4.9 Parameters (PK Parameter Analysis Set) Table 14-9.2.9. Summary of ABP 798 PK Parameters (PK Parameter Analysis Set) Table 14-9.2.10. Summary of Rituximab (US) PK Parameters (PK Parameter Analysis Set) Table 14-9.2.11. Summary of Rituximab (EU) PK Parameters (PK Parameter Analysis Set) Summary of Statistical Assessment of PK Parameters (PK Table 14-9.3.1.1. Parameter Analysis Set) Summary of Statistical Assessment of PK Parameters for Negative Table 14-9.3.1.2. Binding ADA Status Subgroup (PK Parameter Analysis Set) Table 14-9.3.1.3. Summary of Statistical Assessment of PK Parameters for Negative Neutralizing ADA Status Subgroup (PK Parameter Analysis Set) Table 14-9.3.1.4. Summary of Statistical Assessment of PK Parameters without Covariates (PK Parameter Analysis Set) Summary of Statistical Assessment of PK Parameters (Per Table 14-9.3.2. Protocol PK Parameter Analysis Set) 14.10 **Immunogenicity Data Table** Anti-drug Antibodies Summary Results by Treatment- Day 1 Table 14-10.1.1. Until 1<sup>st</sup> Infusion of the 2nd Dose (ADA Analysis Set)



Statistical Analysis Plan Sponsor: Amgen Inc. Protocol No: 20130108 10-December-2018/ Version 2.0 Anti-drug Antibodies Summary Results by Treatment- Entire Table 14-10.1.2. Study (ADA Analysis Set) 14.11 **Pharmacodynamics** Table 14-11.1.1. Pharmacodynamics Results by Visit (Full Analysis Set) Table 14-11.2. Analysis of CD19+ Complete Depletion by Visit (Full Analysis Set) Table 14-11.3. Duration of CD19+ Complete Depletion (Full Analysis Set) 16.1 **Study Information Listings** Listing of Unique Manufacturing Lot Numbers Listing 16-1.6.1. Listing 16-1.6.2. Listing of Subjects Receiving Investigational Product – Subject Listing of Manufacturing Lot Numbers (Safety Analysis Set) Listing 16-1.7. Randomization Assignments (All Randomized Subjects) 16.2 **Subject Data Listings** Listing 16-2.1.1. Subject Listing of Disposition (All Randomized Subjects) Listing 16-2.1.2. Subject Listing of Screen Failures (All Screened Subjects) Listing 16-2.2. Important Protocol Deviations (Full Analysis Set) Listing 16-2.3. Inclusion/Exclusion Criteria Protocol Deviations (Full Analysis Set) Listing 16-2.4. Deviation/Exclusion From Analysis Populations (All Randomized Subjects) Listing 16-2.5. Investigational Product Administration (Safety Analysis Set) Listing 16-2.6.1. Blood Sampling Times and Serum ABP 798 and Rituximab Concentration Data (PK Concentration Analysis Set) Listing 16-Individual PK Parameters from PK Analysis of ABP 798 (PK 2.6.2.1.1 Parameter Analysis Set) Individual PK Parameters from PK Analysis of Rituximab (US) Listing 16-2.6.2.2.1 (PK Parameter Analysis Set) Listing 16-Individual PK Parameters from PK Analysis of Rituximab (EU) 2.6.2.3.1 (PK Parameter Analysis Set)

2.6.2.3.1 (PK Parameter Analysis Set)

Listing 16-2.7.1. Subjects Who Experienced Treatment-emergent Adverse Events Leading to Discontinuation of Study IP/Study (Safety Analysis Set)

Listing 16-2.7.2. Subjects with Treatment-emergent Adverse Events with Fatal Outcome (Safety Analysis Set)



Sponsor: Amgen Inc.

Statistical Analysis Plan

Protocol No: 20130108

10-December-2018/ Version 2.0

Listing 16-2.7.3.Subjects Who Experienced Serious Treatment-emergent Adverse<br/>Events (Safety Analysis Set)Listing 16-2.8.1.Subjects Who Experienced a Grade ≥3 Hematology Result (Safety<br/>Analysis Set)Listing 16-2.8.2.Subjects Who Experienced a Grade≥3 Serum Chemistry Result<br/>(Safety Analysis Set)Listing 16-2.8.3.Subject Binding and Neutralizing Antibody Classification –<br/>Through Entire Study (ADA Analysis Set)Listing 16-2-8.4.On-study Procedure (Safety Analysis Set)

#### SUPPORTIVE SAS OUTPUT APPENDICES

| Appendix 1 | Statistical Output of Table 14-4.1.1: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline at Week 24<br>– Primary Analysis (Full Analysis Set) |
|---|---|
| Appendix 2 | Statistical Output of Table 14-4.1.2: Analysis of DAS28-CRP Change From Baseline at Week 24 – Sensitivity Analysis (Full Analysis Set) |
| Appendix 3 | Statistical Output of Table 14-4.1.3.1: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline by Visit –<br>Day 1 Through Week 24 (Full Analysis Set) |
| Appendix 4 | Statistical Output of Table 14-4.1.3.2: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline by Visit –<br>Day 1 Through Week 24 (Per Protocol Analysis Set) |
| Appendix 5 | Statistical Output of Table 14-4.1.4.1: Analysis of DAS28-CRP Change From Baseline by Visit – Day 1 Through End of Study (Full Analysis Set) |
| Appendix 6 | Statistical Output of Table 14-4.1.4.2: Analysis of DAS28-CRP Change From Baseline by Visit – Day 1 Through End of Study (Full Analysis Set – Subgroup who received the 1st infusion of the 2nd dose at week 24) |
| Appendix 7 | Statistical Output of Table 14-4.1.6: Tipping Point Analysis Results for Mean Difference of DAS28-CRP Change From Baseline at Week 24 for ABP 798 vs Rituximab with 90% Confidence Interval (Full Analysis Set) |
| Appendix 8 | Statistical Output of Table 14-4.1.7: Repeated Measures<br>Analysis with Additional Selective Covariates for DAS28-<br>CRP Change From Baseline at Week 24 (Full Analysis Set) |



| Appendix 9 | Statistical Output of Table 14-4.2.1: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline by Age<br>Subgroup - Day 1 Through Week 24 (Full Analysis Set) |
|---|---|
| Appendix 10 | Statistical Output of Table 14-4.2.2: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline by Race<br>Subgroup – Day 1 Through Week 24 (Full Analysis Set) |
| Appendix 11 | Statistical Output of Table 14-4.2.3: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline by Gender<br>Subgroup – Day 1 Through Week 24 (Full Analysis Set) |
| Appendix 12 | Statistical Output of Table 14-4.2.5: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline by Binding<br>Anti-drug Antibodies Status Subgroup – Day 1 Through<br>Week 24 (Full Analysis Set) |
| Appendix 13 | Statistical Output of Table 14-4.2.6: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline by<br>Neutralizing Anti-drug Antibodies Status Subgroup – Day 1<br>Through Week 24 (Full Analysis Set) |
| Appendix 14 | Statistical Output of Table 14-4.2.7: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline by Baseline<br>Oral Corticosteroid Use Subgroup – Day 1 Through Week<br>24 (Full Analysis Set) |
| Appendix 15 | Statistical Output of Table 14-4.3.1: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline by<br>Geographic Region Subgroup – Day 1 Through Week 24<br>(Full Analysis Set) |
| Appendix 16 | Statistical Output of Table 14-4.3.2: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline by<br>Seropositivity Subgroup – Day 1 Through Week 24 (Full<br>Analysis Set) |
| Appendix 17 | Statistical Output of Table 14-4.3.3: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline by Prior<br>Biologics Use Subgroup – Day 1 Through Week 24 (Full<br>Analysis Set) |
| Appendix 18 | Statistical Output of Table 14-4.5.1.1: Repeated Measures<br>Analysis of ACR20 by Visit – Day 1 Through Week 24 (Full<br>Analysis Set) |
| Appendix 19 | Statistical Output of Table 14-4.5.1.2: Repeated Measures<br>Analysis of ACR20 by Visit – Day 1 Through Week 24 (Per<br>Protocol Analysis Set) |



| Appendix 20 | Statistical Output of Table 14-4.5.2.1: Analysis of ACR20 by Visit – Day 1 Through End of Study (Full Analysis Set) |
|---|---|
| Appendix 21 | Statistical Output of Table 14-4.5.2.2: Analysis of ACR20 by Visit – Day 1 Through End of Study (Full Analysis Set – Subgroup who received the 1st infusion of the 2nd dose at week 24) |
| Appendix 22 | Statistical Output of Table 14-4.5.3.1: Repeated Measures<br>Analysis of Hybrid ACR by Visit – Day 1 Through Week 24<br>(Full Analysis Set) |
| Appendix 23 | Statistical Output of Table 14-4.5.3.2: Repeated Measures<br>Analysis of Hybrid ACR by Visit – Day 1 Through Week 24<br>(Per Protocol Set) |
| Appendix 24 | Statistical Output of Table 14-4.5.3.3: Analysis of Hybrid ACR by Visit – Day 1 Through End of Study (Full Analysis Set) |
| Appendix 25 | Statistical Output of Table 14-4.5.3.4: Analysis of Hybrid ACR by Visit – Day 1 Through End of Study (Full Analysis Set – Subgroup who received the 1st infusion of the 2nd dose at week 24) |
| Appendix 26 | Statistical Output of Table 14-4.6.1: Repeated Measures<br>Analysis of ACR50 by Visit – Day 1 Through Week 24 (Full<br>Analysis Set) |
| Appendix 27 | Statistical Output of Table 14-4.6.2.1: Analysis of ACR50 by Visit – Day 1 Through End of Study (Full Analysis Set) |
| Appendix 28 | Statistical Output of Table 14-4.6.2.2: Analysis of ACR50 by Visit – Day 1 Through End of Study (Full Analysis Set – Subgroup who received the 1st infusion of the 2nd dose at week 24) |
| Appendix 29 | Statistical Output of Table 14-4.7.1: Repeated Measures<br>Analysis of ACR70 by Visit – Day 1 Through Week 24 (Full<br>Analysis Set) |
| Appendix 30 | Statistical Output of Table 14-4.7.2.1: Analysis of ACR70 by Visit – Day 1 Through End of Study (Full Analysis Set) |
| Appendix 31 | Statistical Output of Table 14-4.7.2.2: Analysis of ACR70 by Visit – Day 1 Through End of Study (Full Analysis Set–Subgroup who received the 1st infusion of the 2nd dose at week 24) |
| Appendix 32 | Statistical Output of Table 14-4.10.1.1: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline at Week 24 |



| 20120100 | |
|---|---|
| | Comparing ABP 798 with Pooled Rituximab (Full Analysis Set) |
| Appendix 33 | Statistical Output of Table 14-4.10.1.2: Analysis of DAS28-CRP Change From Baseline (ANCOVA) at Week 24 Comparing ABP 798 with Pooled Rituximab (Full Analysis Set) |
| Appendix 34 | Statistical Output of Table 14-4.10.1.3.1: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline Comparing<br>ABP 798 with Pooled Rituximab by Visit – Day 1<br>ThroughWeek 24 (Full Analysis Set) |
| Appendix 35 | Statistical Output of Table 14-4.10.1.3.2: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline Comparing<br>ABP 798 with Pooled Rituximab by Visit – Day 1 Through<br>Week 24 (Per Protocol Analysis Set) |
| Appendix 36 | Statistical Output of Table 14-4.10.1.4.1: Analysis of DAS28-CRP Change From Baseline (ANCOVA) Comparing ABP 798 with Pooled Rituximab by Visit – Day 1 Through End of Study (Full Analysis Set) |
| Appendix 37 | Statistical Output of Table 14-4.10.1.4.2: Analysis of DAS28-CRP Change From Baseline (ANCOVA) Comparing ABP 798 with Pooled Rituximab by Visit – Day 1 Through End of Study (Per Protocol Set) |
| Appendix 38 | Statistical Output of Table 14-4.10.1.6: Tipping Point Analysis Results for Mean Difference of DAS28-CRP Change From Baseline at Week 24 for ABP 798 vs Pooled Rituximab with 90% Confidence Interval (Full Analysis Set) |
| Appendix 39 | Statistical Output of Table 14-4.10.1.7: Repeated Measures<br>Analysis with Additional Selective Covariates for DAS28-<br>CRP Change From Baseline at Week 24 Comparing ABP<br>798 with Pooled Rituximab (Full Analysis Set) |
| Appendix 40 | Statistical Output of Table 14-4.10.5.1: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline Comparing<br>ABP 798 with Pooled Rituximab by Age Subgroup - Day 1<br>Through Week 24 (Full Analysis Set) |
| Appendix 41 | Statistical Output of Table 14-4.10.5.2: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline Comparing<br>ABP 798 with Pooled Rituximab by Race Subgroup – Day 1<br>Through Week 24 (Full Analysis Set) |
| Appendix 42 | Statistical Output of Table 14-4.10.5.3: Repeated Measures Analysis of DAS28-CRP Change From Baseline Comparing |

Statistical Analysis Plan Sponsor: Amgen Inc. 10-December-2018/ Version 2.0 Protocol No: 20130108

| 20120100 | 10 D 000 movi 2010/ |
|---|---|
| | ABP 798 with Pooled Rituximab by Gender Subgroup – Day<br>1 Through Week 24 (Full Analysis Set) |
| Appendix 43 | Statistical Output of Table 14-4.10.5.5: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline Comparing<br>ABP 798 with Pooled Rituximab by Binding Anti-drug<br>Antibodies Status Subgroup – Day 1 Through Week 24 (Full<br>Analysis Set) |
| Appendix 44 | Statistical Output of Table 14-4.10.5.6: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline Comparing<br>ABP 798 with Pooled Rituximab by Neutralizing Anti-drug<br>Antibodies Status Subgroup – Day 1 Through Week 24 (Full<br>Analysis Set) |
| Appendix 45 | Statistical Output of Table 14-4.10.5.7: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline Comparing<br>ABP 798 with Pooled Rituximab by Baseline Oral<br>Corticosteroid Use Subgroup – Day 1 Through Week 24<br>(Full Analysis Set) |
| Appendix 46 | Statistical Output of Table 14-4.10.6.1: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline Comparing<br>ABP 798 with Pooled Rituximab by Geographic Region<br>Subgroup – Day 1 Through Week 24 (Full Analysis Set) |
| Appendix 47 | Statistical Output of Table 14-4.10.6.2: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline Comparing<br>ABP 798 with Pooled Rituximab by Seropositivity Subgroup<br>– Day 1 Through Week 24 (Full Analysis Set) |
| Appendix 48 | Statistical Output of Table 14-4.10.6.3: Repeated Measures<br>Analysis of DAS28-CRP Change From Baseline Comparing<br>ABP 798 with Pooled Rituximab by Prior Biologics Use<br>Subgroup – Day 1 Through Week 24 (Full Analysis Set) |
| Appendix 49 | Statistical Output of Table 14-4.11.5.1.1: Repeated Measures<br>Analysis of ACR20 Comparing ABP 798 with Pooled<br>Rituximab by Visit – Day 1 Through Week 24 (Full<br>Analysis Set) |
| Appendix 50 | Statistical Output of Table 14-4.11.5.1.2: Repeated Measures<br>Analysis of ACR20 Comparing ABP 798 with Pooled<br>Rituximab by Visit – Day 1 Through Week 24 (Per Protocol<br>Analysis Set) |
| Appendix 51 | Statistical Output of Table 14-4.12.1.1: Repeated Measures<br>Analysis of Hybrid ACR Comparing ABP 798 with Pooled<br>Rituximab by Visit – Day 1 Through Week 24 (Full<br>Analysis Set) |



Statistical Analysis Plan Sponsor: Amgen Inc. 10-December-2018/ Version 2.0 Protocol No: 20130108

| Appendix 52 | Statistical Output of Table 14-4.12.1.2: Repeated Measures<br>Analysis of Hybrid ACR Comparing ABP 798 with Pooled<br>Rituximab by Visit – Day 1 Through Week 24 (Per Protocol<br>Analysis Set) |
|---|---|
| Appendix 53 | Statistical Output of Table 14-4.13.1: Repeated Measures<br>Analysis of ACR50 Comparing ABP 798 with Pooled<br>Rituximab by Visit – Day 1 Through Week 24 (Full<br>Analysis Set) |
| Appendix 54 | Statistical Output of Table 14-4.14.1: Repeated Measures<br>Analysis of ACR70 Comparing ABP 798 with Pooled<br>Rituximab by Visit – Day 1 Through Week 24 (Full<br>Analysis Set) |
| Appendix 55 | Statistical Output of Table 14-6.5.1.1: Overall Events of Interest Treatment-emergent Adverse Events by Treatment – Day 1 Until 1st Infusion of 2nd Dose (Safety Analysis Set) |
| Appendix 56 | Statistical Output of Table 14-6.7.1: Exposure Adjusted Incidence Rate for Treatment-emergent Adverse Events by Preferred Term and Treatment - Day 1 Through End of Study (Safety Analysis Set) |
| Appendix 57 | Statistical Output of Table 14-6.7.2: Exposure Adjusted Incidence Rate for Treatment-emergent Adverse Events of Interest by Treatment – Day 1 Through End of Study (Safety Analysis Set) |
| Appendix 58 | Statistical Output of Table 14-9.3.1.1: Summary of Statistical Assessment of PK Parameters (PK Parameter Analysis Set) |
| Appendix 59 | Statistical Output of Table 14-9.3.1.2: Summary of Statistical Assessment of PK Parameters for Negative Binding ADA Status Subgroup (PK Parameter Analysis Set) |
| Appendix 60 | Statistical Output of Table 14-9.3.1.3: Summary of<br>Statistical Assessment of PK Parameters for Negative<br>Neutralizing ADA Status Subgroup (PK Parameter Analysis<br>Set) |
| Appendix 61 | Statistical Output of Table 14-9.3.1.4: Summary of Statistical Assessment of PK Parameters without Covariates (PK Parameter Analysis Set) |
| Appendix 62 | Statistical Output of Table 14-9.3.2: Summary of Statistical Assessment of PK Parameters (Per Protocol PK Parameter Analysis Set) |




Appendix 63 Statistical Output of Table 14-11.2: Analysis of CD19+

Complete Depletion by Visit (Full Analysis Set)

Appendix 64 Statistical Output of Table 14-11.3: Duration of CD19+

Complete Depletion (Full Analysis Set)




# APPENDIX 7 SHELLS FOR POST-TEXT TABLES, FIGURES, AND LISTINGS

See associated TFL shell document.